CLINICAL TRIAL: NCT01146652
Title: A Multi-center, Uncontrolled Extension Study Evaluating Efficacy and Safety of SAR153191 in Patients With Active Rheumatoid Arthritis (RA)
Brief Title: Long Term Evaluation of Sarilumab in Rheumatoid Arthritis Patients (SARIL-RA-EXTEND)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LTS11210; 2010-019262-86 (EudraCT Number)
Record Dates: First submitted 2010-06-15; First posted 2010-06-17 (Estimated); Results first posted 2022-01-24 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — sarilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sarilumab + Disease Modifying Anti-Rheumatic Drugs (DMARD) (Experimental): Participants who completed any of initial studies:Part A or B of EFC11072, ACT11575, EFC10832 or SFY13370 were enrolled in LTS11210 and received sarilumab 150 milligrams (mg) subcutaneously (SC) once weekly (qw). Dose could be reduced to 150 mg every 2 weeks (q2w) due to neutropenia, thrombocytopenia or increase in liver enzymes (alanine aminotransferase [ALT]). After dose regimens selection for Phase 3 studies (150 mg q2w and 200 mg q2w), participants already receiving 150 mg qw were switched to sarilumab 200 mg q2w. Treatment duration per participant was at least 264 weeks from first study drug administration in LTS11210. Participants continued to be treated beyond 264 weeks until sarilumab was commercially available in their respective countries or until 2020, at the latest (maximum duration: 523 weeks). Participants who were already taking concomitant non-biologic DMARDs in initial study continued stable dose of one or combination of conventional synthetic DMARDs they were taking.
  Interventions: Drug: SAR153191 (REGN88)
- Sarilumab monotherapy (Experimental): Participants who completed study EFC13752 were enrolled in LTS11210 and received sarilumab 200 mg q2w. Dose could be reduced to 150 mg q2w due to neutropenia, thrombocytopenia or increase in liver enzymes (ALT). Treatment duration per participant was at least 264 weeks from first study drug administration in LTS11210. Participants continued to be treated beyond 264 weeks until sarilumab was commercially available in their respective countries or until 2020, at the latest (maximum duration: 523 weeks).
  Interventions: Drug: SAR153191 (REGN88)

INTERVENTIONS:
Drug: SAR153191 (REGN88) — Pharmaceutical form: solution
  Route of administration: subcutaneous

SUMMARY:
Main Study:

Primary Objective:

Assess the long term safety of sarilumab in participants with rheumatoid arthritis (RA).

Secondary Objective:

Assess the long term efficacy of sarilumab in participants with RA.

Sub-Study:

This phase 3, open label sub-study was aimed to assess the usability of PFS-S when used by participants with moderate or severe RA, or their professional or non-professional healthcare providers in an unsupervised real-world situation. To mimic the real-world practice, the sub-study was incorporated into the LTS11210 study without additional visits compared to the scheduled visits in the main study. The duration of this sub-study was 12 weeks.

DETAILED DESCRIPTION:
The maximum duration of the study was up to 523 weeks:

* Up to 1-week of screening, if any.
* At least 264 weeks of open label treatment phase and up to 516 weeks as maximum.
* 6-week post-treatment follow-up as required per protocol.

ELIGIBILITY:
Inclusion criteria :

Main study:

Participants with RA who were previously randomized in the sarilumab RA clinical program: e.g., the EFC11072 study, ACT11575 study, EFC10832 study, SFY13370, and EFC13752 study.

Sub-study:

Participants enrolled in the LTS11210 study who were receiving either sarilumab 200mg q2w PFS or sarilumab 150mg q2w PFS and who were able and willing to participate in this sub-study.

Participants who had been enrolled in the main study for at least 24 weeks. Participants must sign a sub-study written informed consent prior to any sub-study related procedure.

Exclusion criteria:

Main study:

Participants with any adverse event (AE) led to permanent study drug discontinuation from a prior study.

Participants with an abnormality(ies) or AEs that per investigator judgment would adversely affect participation of the participant in the study.

Sub-study: There are no additional exclusion criteria to those defined in main study.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2023 (Actual)
Dates: Start 2010-06-21 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences and Operations, Study Director — Sanofi
Locations (335):
- United States (75):
  - Investigational Site Number 840070, Anniston, Alabama
  - Investigational Site Number 840138, Birmingham, Alabama
  - Investigational Site Number 840152, Huntsville, Alabama
  - Investigational Site Number 840072, Gilbert, Arizona
  - Investigational Site Number 840141, Glendale, Arizona
  - Investigational Site Number 840134, Fullerton, California
  - Investigational Site Number 840008, La Jolla, California
  - Investigational Site Number 840135, San Diego, California
  - Investigational Site Number 840021, Santa Maria, California
  - Investigational Site Number 840100, Stanford, California
  - Investigational Site Number 840049, Upland, California
  - Investigational Site Number 840151, Colorado Springs, Colorado
  - Investigational Site Number 840130, Lewes, Delaware
  - Investigational Site Number 840153, Aventura, Florida
  - Investigational Site Number 840050, Clearwater, Florida
  - Investigational Site Number 840033, Fort Lauderdale, Florida
  - Investigational Site Number 840041, Gainesville, Florida
  - Investigational Site Number 840067, Jupiter, Florida
  - Investigational Site Number 840048, Miami, Florida
  - Investigational Site Number 840024, Naples, Florida
  - Investigational Site Number 840006, Orlando, Florida
  - Investigational Site Number 840128, Ormond Beach, Florida
  - Investigational Site Number 840063, Palm Harbor, Florida
  - Investigational Site Number 840155, Palm Harbor, Florida
  - Investigational Site Number 840060, Sarasota, Florida
  - Investigational Site Number 840140, Tampa, Florida
  - Investigational Site Number 840126, Vero Beach, Florida
  - Investigational Site Number 840003, Atlanta, Georgia
  - Investigational Site Number 840028, Decatur, Georgia
  - Investigational Site Number 840027, Marietta, Georgia
  - Investigational Site Number 840018, Idaho Falls, Idaho
  - Investigational Site Number 840046, Chicago, Illinois
  - Investigational Site Number 840052, Kansas City, Kansas
  - Investigational Site Number 840230, Elizabethtown, Kentucky
  - Investigational Site Number 840015, Lexington, Kentucky
  - Investigational Site Number 840120, Baton Rouge, Louisiana
  - Investigational Site Number 840109, Lake Charles, Louisiana
  - Investigational Site Number 840055, Frederick, Maryland
  - Investigational Site Number 840013, Wheaton, Maryland
  - Investigational Site Number 840154, Boston, Massachusetts
  - Investigational Site Number 840150, Lansing, Michigan
  - Investigational Site Number 840137, Saint Clair Shores, Michigan
  - Investigational Site Number 840112, Lincoln, Nebraska
  - Investigational Site Number 840026, Freehold, New Jersey
  - Investigational Site Number 840115, Lake Success, New York
  - Investigational Site Number 840056, New York, New York
  - Investigational Site Number 840043, New York, New York
  - Investigational Site Number 840106, Orchard Park, New York
  - Investigational Site Number 840118, Smithtown, New York
  - Investigational Site Number 840116, Wilmington, North Carolina
  - Investigational Site Number 840233, Minot, North Dakota
  - Investigational Site Number 840002, Oklahoma City, Oklahoma
  - Investigational Site Number 840127, Oklahoma City, Oklahoma
  - Investigational Site Number 840011, Tulsa, Oklahoma
  - Investigational Site Number 840065, Tulsa, Oklahoma
  - Investigational Site Number 840010, Bethlehem, Pennsylvania
  - Investigational Site Number 840009, Duncansville, Pennsylvania
  - Investigational Site Number 840062, Reading, Pennsylvania
  - Investigational Site Number 840058, Columbia, South Carolina
  - Investigational Site Number 840016, North Charleston, South Carolina
  - Investigational Site Number 840025, Jackson, Tennessee
  - Investigational Site Number 840059, Memphis, Tennessee
  - Investigational Site Number 840032, Amarillo, Texas
  - Investigational Site Number 840038, Austin, Texas
  - Investigational Site Number 840001, Dallas, Texas
  - Investigational Site Number 840022, Dallas, Texas
  - Investigational Site Number 840012, Dallas, Texas
  - Investigational Site Number 840129, Houston, Texas
  - Investigational Site Number 840069, Lubbock, Texas
  - Investigational Site Number 840074, Mesquite, Texas
  - Investigational Site Number 840020, Nassau Bay, Texas
  - Investigational Site Number 840103, San Antonio, Texas
  - Investigational Site Number 840036, Spokane, Washington
  - Investigational Site Number 840061, Tacoma, Washington
  - Investigational Site Number 840124, Clarksburg, West Virginia
- Argentina (18):
  - Investigational Site Number 032006, Caba
  - Investigational Site Number 032007, Caba
  - Investigational Site Number 032008, Caba
  - Investigational Site Number 032019, Capital Federal
  - Investigational Site Number 032016, Capital Federal
  - Investigational Site Number 032002, Córdoba
  - Investigational Site Number 032020, Córdoba
  - Investigational Site Number 032003, Córdoba
  - Investigational Site Number 032017, La Plata
  - Investigational Site Number 032012, Mar del Plata
  - Investigational Site Number 032011, Quilmes
  - Investigational Site Number 032010, Ramos Mejía
  - Investigational Site Number 032001, Rosario
  - Investigational Site Number 032013, Rosario
  - Investigational Site Number 032015, San Fernando
  - Investigational Site Number 032005, San Miguel de Tucumán
  - Investigational Site Number 032004, San Miguel de Tucumán
  - Investigational Site Number 032009, Zárate
- Australia (7):
  - Investigational Site Number 036003, Camperdown
  - Investigational Site Number 036012, Fitzroy
  - Investigational Site Number 036010, Garran
  - Investigational Site Number 036004, Heidelberg West
  - Investigational Site Number 036001, Maroochydore
  - Investigational Site Number 036014, Victoria Park
  - Investigational Site Number 036007, Woodville
- Investigational Site Number 040001, Graz, Austria
- Belarus (2):
  - Investigational Site Number 112002, Minsk
  - Investigational Site Number 112001, Minsk
- Investigational Site Number 056010, Leuven, Belgium
- Brazil (10):
  - Investigational Site Number 076001, Curitiba
  - Investigational Site Number 076006, Goiânia
  - Investigational Site Number 076010, Juiz de Fora
  - Investigational Site Number 076004, Porto Alegre
  - Investigational Site Number 076005, Rio de Janeiro
  - Investigational Site Number 076015, Rio de Janeiro
  - Investigational Site Number 076011, Salvador
  - Investigational Site Number 076002, São Paulo
  - Investigational Site Number 076003, São Paulo
  - Investigational Site Number 076013, Vitória
- Canada (6):
  - Investigational Site Number 124003, Mississauga
  - Investigational Site Number 124002, St. Catharines
  - Investigational Site Number 124005, Toronto
  - Investigational Site Number 124009, Trois-Rivières
  - Investigational Site Number 124104, Victoria
  - Investigational Site Number 124012, Winnipeg
- Chile (13):
  - Investigational Site Number 152005, Osorno
  - Investigational Site Number 152012, Santiago
  - Investigational Site Number 152002, Santiago
  - Investigational Site Number 152011, Santiago
  - Investigational Site Number 152009, Santiago
  - Investigational Site Number 152001, Santiago
  - Investigational Site Number 152013, Santiago
  - Investigational Site Number 152008, Santiago
  - Investigational Site Number 152014, Talca
  - Investigational Site Number 152015, Temuco IX Region
  - Investigational Site Number 152004, Valdivia
  - Investigational Site Number 152007, Viña del Mar
  - Investigational Site Number 152006, Viña del Mar
- Colombia (8):
  - Investigational Site Number 170005, Barranquilla
  - Investigational Site Number 170004, Barranquilla
  - Investigational Site Number 170006, Bogotá
  - Investigational Site Number 170001, Bogotá
  - Investigational Site Number 170003, Bogotá
  - Investigational Site Number 170008, Bogotá
  - Investigational Site Number 170007, Bucaramanga
  - Investigational Site Number 170009, Bucaramanga
- Czechia (9):
  - Investigational Site Number 203009, Liberec
  - Investigational Site Number 203004, Ostrava
  - Investigational Site Number 203034, Pardubice
  - Investigational Site Number 203001, Prague
  - Investigational Site Number 203007, Prague
  - Investigational Site Number 203011, Prague
  - Investigational Site Number 203010, Prague
  - Investigational Site Number 203002, Uherské Hradiště
  - Investigational Site Number 203006, Zlín
- Ecuador (3):
  - Investigational Site Number 218003, Cuenca
  - Investigational Site Number 218001, Guayaquil
  - Investigational Site Number 218002, Quito
- Estonia (3):
  - Investigational Site Number 233001, Tallinn
  - Investigational Site Number 233010, Tallinn
  - Investigational Site Number 233002, Tallinn
- Finland (4):
  - Investigational Site Number 246001, Helsinki
  - Investigational Site Number 246002, Hyvinkää
  - Investigational Site Number 246003, Pori
  - Investigational Site Number 246010, Riihimäki
- Germany (15):
  - Investigational Site Number 276011, Bad Nauheim
  - Investigational Site Number 276010, Berlin
  - Investigational Site Number 276007, Berlin
  - Investigational Site Number 276008, Berlin
  - Investigational Site Number 276014, Berlin
  - Investigational Site Number 276018, Deggingen
  - Investigational Site Number 276015, Halle
  - Investigational Site Number 276005, Hamburg
  - Investigational Site Number 276013, Hamburg
  - Investigational Site Number 276001, Herne
  - Investigational Site Number 276016, Leipzig
  - Investigational Site Number 276017, München
  - Investigational Site Number 276021, Osnabrück
  - Investigational Site Number 276020, Tübingen
  - Investigational Site Number 276019, Zerbst
- Greece (3):
  - Investigational Site Number 300002, Heraklion
  - Investigational Site Number 300003, Thessaloniki
  - Investigational Site Number 300005, Thessaloniki
- Guatemala (3):
  - Investigational Site Number 320002, Guatemala City
  - Investigational Site Number 320003, Guatemala City
  - Investigational Site Number 320001, Guatemala City
- Hungary (12):
  - Investigational Site Number 348006, Budapest
  - Investigational Site Number 348014, Budapest
  - Investigational Site Number 348025, Budapest
  - Investigational Site Number 348022, Budapest
  - Investigational Site Number 348010, Debrecen
  - Investigational Site Number 348003, Debrecen
  - Investigational Site Number 348021, Esztergom
  - Investigational Site Number 348013, Győr
  - Investigational Site Number 348005, Sátoraljaújhely
  - Investigational Site Number 348004, Székesfehérvár
  - Investigational Site Number 348009, Szolnok
  - Investigational Site Number 348015, Szombathely
- Israel (4):
  - Investigational Site Number 376001, Haifa
  - Investigational Site Number 376010, Haifa
  - Investigational Site Number 376011, Tel Aviv
  - Investigational Site Number 376002, Tel Litwinsky
- Investigational Site Number 380005, Genova, Italy
- Lithuania (4):
  - Investigational Site Number 440001, Kaunas
  - Investigational Site Number 440006, Klaipėda
  - Investigational Site Number 440002, Vilnius
  - Investigational Site Number 440007, Vilnius
- Malaysia (2):
  - Investigational Site Number 458001, Ipoh
  - Investigational Site Number 458002, Kuching
- Mexico (16):
  - Investigational Site Number 484023, Chihuahua City
  - Investigational Site Number 484008, Durango
  - Investigational Site Number 484018, Guadalajara
  - Investigational Site Number 484002, Guadalajara
  - Investigational Site Number 484035, León
  - Investigational Site Number 484007, Metepec
  - Investigational Site Number 484010, Mexicali
  - Investigational Site Number 484003, Mexico City
  - Investigational Site Number 484009, Mérida
  - Investigational Site Number 484004, Mérida
  - Investigational Site Number 484017, México
  - Investigational Site Number 484001, México, D.F.
  - Investigational Site Number 484019, Monterrey
  - Investigational Site Number 484020, Monterrey
  - Investigational Site Number 484005, Monterrey
  - Investigational Site Number 484021, Querétaro
- Investigational Site Number 528010, Amsterdam, Netherlands
- New Zealand (5):
  - Investigational Site Number 554004, Christchurch
  - Investigational Site Number 554011, Nelson
  - Investigational Site Number 554007, Otahuhu
  - Investigational Site Number 554002, Rotorua
  - Investigational Site Number 554001, Timaru
- Peru (9):
  - Investigational Site Number 604001, Lima
  - Investigational Site Number 604010, Lima
  - Investigational Site Number 604008, Lima
  - Investigational Site Number 604009, Lima
  - Investigational Site Number 604006, Lima
  - Investigational Site Number 604012, Lima
  - Investigational Site Number 604013, Lima
  - Investigational Site Number 604007, Lima
  - Investigational Site Number 604005, Lima
- Philippines (2):
  - Investigational Site Number 608003, Cebu City
  - Investigational Site Number 608001, Manila
- Poland (17):
  - Investigational Site Number 616014, Bialystok
  - Investigational Site Number 616002, Bialystok
  - Investigational Site Number 616003, Bialystok
  - Investigational Site Number 616019, Bydgoszcz
  - Investigational Site Number 616054, Bytom
  - Investigational Site Number 616015, Elblag
  - Investigational Site Number 616001, Krakow
  - Investigational Site Number 616005, Lublin
  - Investigational Site Number 616030, Lublin
  - Investigational Site Number 616018, Poznan
  - Investigational Site Number 616016, Szczecin
  - Investigational Site Number 616006, Torun
  - Investigational Site Number 616031, Warsaw
  - Investigational Site Number 616004, Warsaw
  - Investigational Site Number 616017, Warsaw
  - Investigational Site Number 616020, Wroclaw
  - Investigational Site Number 616012, Wroclaw
- Investigational Site Number 620002, Lisbon, Portugal
- Romania (7):
  - Investigational Site Number 642006, Brăila
  - Investigational Site Number 642021, Bucharest
  - Investigational Site Number 642001, Bucharest
  - Investigational Site Number 642010, Bucharest
  - Investigational Site Number 642020, Bucharest
  - Investigational Site Number 642002, Bucharest
  - Investigational Site Number 642005, Galati
- Russia (19):
  - Investigational Site Number 643006, Kemerovo
  - Investigational Site Number 643017, Kemerovo
  - Investigational Site Number 643020, Moscow
  - Investigational Site Number 643001, Moscow
  - Investigational Site Number 643002, Moscow
  - Investigational Site Number 643021, Moscow
  - Investigational Site Number 643004, Moscow
  - Investigational Site Number 643012, Moscow
  - Investigational Site Number 643031, Moscow
  - Investigational Site Number 643030, Moscow
  - Investigational Site Number 643009, Novosibirsk
  - Investigational Site Number 643016, Ryazan
  - Investigational Site Number 643007, Saint Petersburg
  - Investigational Site Number 643032, Saint Petersburg
  - Investigational Site Number 643008, Saint Petersburg
  - Investigational Site Number 643014, Saint Petersburg
  - Investigational Site Number 643010, Samara
  - Investigational Site Number 643011, Saratov
  - Investigational Site Number 643013, Ufa
- South Africa (10):
  - Investigational Site Number 710011, Cape Town
  - Investigational Site Number 710007, Cape Town
  - Investigational Site Number 710009, Cape Town
  - Investigational Site Number 710003, Durban
  - Investigational Site Number 710002, Durban
  - Investigational Site Number 710001, Johannesburg
  - Investigational Site Number 710004, Kempton Park
  - Investigational Site Number 710005, Pretoria
  - Investigational Site Number 710006, Pretoria
  - Investigational Site Number 710010, Stellenbosch
- South Korea (14):
  - Investigational Site Number 410014, Anyang-si
  - Investigational Site Number 410006, Busan
  - Investigational Site Number 410004, Daegu
  - Investigational Site Number 410017, Daejeon
  - Investigational Site Number 410005, Daejeon
  - Investigational Site Number 410010, Gwangju
  - Investigational Site Number 410001, Incheon
  - Investigational Site Number 410009, Incheon
  - Investigational Site Number 410011, Jeonju
  - Investigational Site Number 410007, Seoul
  - Investigational Site Number 410012, Seoul
  - Investigational Site Number 410016, Seoul
  - Investigational Site Number 410003, Seoul
  - Investigational Site Number 410008, Suwon
- Spain (10):
  - Investigational Site Number 724009, A Coruña
  - Investigational Site Number 724016, Barakaldo
  - Investigational Site Number 724015, Barcelona
  - Investigational Site Number 724014, Cadiz
  - Investigational Site Number 724001, Málaga
  - Investigational Site Number 724011, Sabadell
  - Investigational Site Number 724012, Santiago de Compostela
  - Investigational Site Number 724013, Santiago de Compostela
  - Investigational Site Number 724022, Seville
  - Investigational Site Number 724007, Seville
- Investigational Site Number 752002, Uppsala, Sweden
- Taiwan (2):
  - Investigational Site Number 158006, Taichung
  - Investigational Site Number 158002, Taoyuan
- Thailand (2):
  - Investigational Site Number 764001, Bangkok
  - Investigational Site Number 764003, Bangkok
- Investigational Site Number 792008, Gaziantep, Turkey (Türkiye)
- Ukraine (10):
  - Investigational Site Number 804003, Dnipro
  - Investigational Site Number 804010, Kharkiv
  - Investigational Site Number 804013, Kharkiv
  - Investigational Site Number 804014, Kyiv
  - Investigational Site Number 804004, Kyiv
  - Investigational Site Number 804027, Kyiv
  - Investigational Site Number 804005, Lviv
  - Investigational Site Number 804006, Simferopol
  - Investigational Site Number 804011, Vinnytsia
  - Investigational Site Number 804009, Zaporizhzhya
- United Kingdom (4):
  - Investigational Site Number 826004, Doncaster
  - Investigational Site Number 826006, Edinburgh
  - Investigational Site Number 826002, Leytonstone
  - Investigational Site Number 826005, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Burmester GR, Strand V, Kivitz AJ, Hu CC, Wang S, van Hoogstraten H, Klier GL, Fleischmann R. Long-term safety and efficacy of sarilumab with or without background csDMARDs in rheumatoid arthritis. Rheumatology (Oxford). 2023 Oct 3;62(10):3268-3279. doi: 10.1093/rheumatology/kead062. PMID 36727470
- [Derived] Choy E, Bykerk V, Lee YC, van Hoogstraten H, Ford K, Praestgaard A, Perrot S, Pope J, Sebba A. Disproportionate articular pain is a frequent phenomenon in rheumatoid arthritis and responds to treatment with sarilumab. Rheumatology (Oxford). 2023 Jul 5;62(7):2386-2393. doi: 10.1093/rheumatology/keac659. PMID 36413080
- [Derived] Fleischmann R, Genovese MC, Maslova K, Leher H, Praestgaard A, Burmester GR. Long-term safety and efficacy of sarilumab over 5 years in patients with rheumatoid arthritis refractory to TNF inhibitors. Rheumatology (Oxford). 2021 Nov 3;60(11):4991-5001. doi: 10.1093/rheumatology/keab355. PMID 33871596
- [Derived] Emery P, van Hoogstraten H, Thangavelu K, Mangan E, St John G, Verschueren P. Subcutaneous Sarilumab in Patients With Rheumatoid Arthritis who Previously Received Subcutaneous Sarilumab or Intravenous Tocilizumab: An Open-Label Extension of a Randomized Clinical Trial. ACR Open Rheumatol. 2020 Nov;2(11):672-680. doi: 10.1002/acr2.11188. Epub 2020 Nov 8. PMID 33164349
- [Derived] Genovese MC, van der Heijde D, Lin Y, St John G, Wang S, van Hoogstraten H, Gomez-Reino JJ, Kivitz A, Maldonado-Cocco JA, Seriolo B, Stanislav M, Burmester GR. Long-term safety and efficacy of sarilumab plus methotrexate on disease activity, physical function and radiographic progression: 5 years of sarilumab plus methotrexate treatment. RMD Open. 2019 Aug 1;5(2):e000887. doi: 10.1136/rmdopen-2018-000887. eCollection 2019. PMID 31452928

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed any of studies EFC11072 (NCT01061736), ACT11575 ( NCT01217814), EFC10832 (NCT01709578), SFY13370 (NCT01768572), EFC13752 (NCT02121210) were eligible for enrollment in LTS11210 (named as main study). A total of 2023 participants were enrolled between 21 June 2010 and 04 May 2015. From Week 24 of LTS11210, willing participants were enrolled in a 12-week sub-study (part of main study only) to assess usability of pre-filled syringe with safety system (PFS-S).
Pre-assignment Details: Participants had been exposed to sarilumab for 12 weeks if they were initially randomized in EFC11072 Part A or ACT11575; for up to 52 weeks if initially randomized in EFC11072 Part B; for up to 24 weeks if initially randomized in EFC10832; or for 24 weeks if initially randomized in SFY13370 or EFC13752. Participant's end-of-treatment visit in initial study corresponded to initial visit in study LTS11210.
Period: Overall Study
Arm/Group | Sarilumab + Disease Modifying Anti-Rheumatic Drugs (DMARD) | Sarilumab Monotherapy
Started | 1912 | 111
Treated | 1910 | 111
Enrolled in the Sub-study (Participants who were eligible and entered sub-study from Week 24 of main study.) | 110 | 14
Discontinued From the Sub-study (Sub-study discontinued participants were included in the discontinuation count of the main study.) | 1 | 2
Switched Back to Main Study (Participants who were willing to switch back to the main study regardless of if they completed the sub-study.) | 108 | 13
Completed | 961 | 66
Not Completed | 951 | 45
Not completed — Adverse Event | 506 | 15
Not completed — Lack of Efficacy | 91 | 7
Not completed — Poor compliance to protocol | 38 | 1
Not completed — Other unspecified reasons | 314 | 22
Not completed — Enrolled but not treated | 2 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all enrolled population.
Arm/Group | Sarilumab + Disease Modifying Anti-Rheumatic Drugs (DMARD) | Sarilumab Monotherapy | Total Title
Number analyzed (Participants) | 1912 | 111 | 2023
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (11.8) | 52.9 (13.1) | 52.2 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1550 | 88 | 1638
  Male | 362 | 23 | 385
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian/White | 1639 | 108 | 1747
  Black | 48 | 1 | 49
  Asian/Oriental | 69 | 1 | 70
  Other | 156 | 1 | 157

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical study participant administered a medicinal product and which did not necessarily have to have a causal relationship with the treatment. An SAE was any untoward medical occurrence at any dose that: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. TEAEs were AEs that developed or worsened or became serious during the TEAE period (defined as the time from the first dose of the investigational medicinal product (IMP) in study LTS11210 to the last dose of the IMP +60 days).
Time Frame: From first dose (i.e., Day 1 of study LTS11210) up to 60 days after last dose (maximum duration: up to 523 weeks)
Population: Analysis was performed on safety population which included all enrolled participants who had received at least one dose of the study treatment in LTS11210.
Measure: Count of Participants; unit: Participants
Arm/Group | Sarilumab + Disease Modifying Anti-Rheumatic Drugs (DMARD) | Sarilumab Monotherapy
Number analyzed (Participants) | 1910 | 111
Participants
  Any TEAE | 1760 | 98
  Any TE SAE | 617 | 27

2. Primary Outcome: Sub-study: Number of Participants Reported Product Technical Complaints (PTC), Product Technical Failures (PTF) and/or Failed Drug Deliveries (FDD) With Pre-filled Syringe With Safety System
Description: A PTF was defined as any product technical complaint (PTC) related to the use of the PFS-S that had a validated technical cause. FDD was defined as participant's failure to administer the full dose at a given attempt. A PTC was defined as any participant- or healthcare provider-reported complaint regarding the use of the PFS-S syringe and collected via the completion of the injection diary. The injection diary comprised specific questions: 1. Were you able to remove the cap? 2. Was the needle safety system activated?, 3. Did the safety system entirely cover the needle, and 4. Was the person who performed the injection the person who was trained by the site staff?, where each question was given the option yes/no. Participants who answered "no" for any of the questions of PTC, had PTF and/or FDD were reported in this outcome measure.
Time Frame: From Week 24 to 36
Population: Analysis was performed on all participants who were enrolled in the sub-study.
Measure: Count of Participants; unit: Participants
Groups:
- PFS-S Sarilumab 150 mg q2w: From Week 24 of main study, eligible participants entered sub-study and received sarilumab 150 mg SC q2w for 12 weeks (i.e., from main study Week 24 to Week 36) using PFS-S.
- PFS-S Sarilumab 200 mg q2w: From Week 24 of main study, eligible participants entered sub-study and received sarilumab 200 mg SC q2w for 12 weeks (i.e., from main study Week 24 to Week 36) using PFS-S.
- PFS-S Sarilumab 200 to 150 mg q2w: From Week 24 of main study, eligible participants entered sub-study and received sarilumab 200 mg SC q2w for 12 weeks (i.e., from main study Week 24 to Week 36) using PF-S. The dose might be reduced to 150 mg q2w due to neutropenia, thrombocytopenia, or an increase in liver enzymes.
Arm/Group | PFS-S Sarilumab 150 mg q2w | PFS-S Sarilumab 200 mg q2w | PFS-S Sarilumab 200 to 150 mg q2w
Number analyzed (Participants) | 25 | 98 | 1
Participants
  PFS-S-associated PTF | 0 | 0 | 0
  PFS-S-associated FDD | 0 | 5 | 0
  PFS-S-associated PTC | 0 | 5 | 0

3. Primary Outcome: Sub-study: Number of Product Technical Complaints - Product Technical Failures With Pre-filled Syringe With Safety System
Description: A PTF was defined as any PTC (defined as any participant- or healthcare provider-reported complaint regarding the use of the PFS-S syringe and collected via the completion of the injection diary) related to the use of the PFS-S that had a validated technical cause. Number of PTF in the participants enrolled in sub-study were reported in this outcome measure.
Time Frame: From Week 24 to 36
Population: Analysis was performed on all participants who were enrolled in the sub-study.
Measure: Number; unit: PTF
Arm/Group | PFS-S Sarilumab 150 mg q2w | PFS-S Sarilumab 200 mg q2w | PFS-S Sarilumab 200 to 150 mg q2w
Number analyzed (Participants) | 25 | 98 | 1
PTF | 0 | 0 | 0

4. Primary Outcome: Sub-study: Number of Failed Drug Deliveries Associated With Pre-filled Syringe With Safety System
Description: FDD was defined as participant's failure to administer the full dose at a given attempt. Number of FDD in the participants enrolled in sub-study were reported in this outcome measure.
Time Frame: From Week 24 to 36
Population: Analysis was performed on all participants who were enrolled in the sub-study.
Measure: Number; unit: FDD
Arm/Group | PFS-S Sarilumab 150 mg q2w | PFS-S Sarilumab 200 mg q2w | PFS-S Sarilumab 200 to 150 mg q2w
Number analyzed (Participants) | 25 | 98 | 1
FDD | 0 | 5 | 0

5. Primary Outcome: Sub-study: Number of Product Technical Complaints With Pre-filled Syringe With Safety System
Description: A PTC was defined as any participant- or healthcare provider-reported complaint regarding the use of the PFS-S syringe and collected via the completion of the injection diary. The injection diary comprised specific questions: 1. Were you able to remove the cap? 2. Was the needle safety system activated?, 3. Did the safety system entirely cover the needle, and 4. Was the person who performed the injection the person who was trained by the site staff?, where each question was given the option yes/no. Number of PTC (based on participant's answer to "no" for any of the questions of PTC) in the participants enrolled in sub-study were reported in this outcome measure.
Time Frame: From Week 24 to 36
Population: Analysis was performed on all participants who were enrolled in the sub-study.
Measure: Number; unit: PTC
Arm/Group | PFS-S Sarilumab 150 mg q2w | PFS-S Sarilumab 200 mg q2w | PFS-S Sarilumab 200 to 150 mg q2w
Number analyzed (Participants) | 25 | 98 | 1
PTC | 0 | 5 | 0

6. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20 (ACR20) Response
Description: ACR20 response: greater than or equal to (>=) 20% improvement in both tender joint count and swollen joint count and, >=20% improvement in at least 3 of the 5 remaining ACR core measures assessments: C-reactive protein [CRP] level (mg/liter [mg/L]); participant's assessment of pain (measured on 0 [no pain] to 100 mm [worst pain] visual analog scale [VAS]); participant's global assessment of disease activity (measured on 0 [no arthritis activity] to 100 mm [maximal arthritis activity] VAS); physician's global assessment of disease activity (measured on 0 [no arthritis activity] to 100 mm [maximal arthritis activity] VAS); participant's assessment of physical function (measured by health assessment questionnaire disability index [HAQ-DI], with scoring range of 0 [better physical function] to 3 [worst physical function]). Higher score indicated worse outcomes.
Time Frame: At Week 0 (post-dose), 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240 and 264 of LTS11210
Population: Analysis was performed on safety population which included participants who had at least 1 dose of study treatment in LTS11210. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure and 'number analyzed' = participants with available data for each specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sarilumab + Disease Modifying Anti-Rheumatic Drugs (DMARD) | Sarilumab Monotherapy
Number analyzed (Participants) | 1898 | 111
percentage of participants
  Week 0 | 69.4 [67.3 to 71.5] | 82.0 [73.6 to 88.6]
  Week 4: number analyzed (Participants) | 1885 | 106
  Week 4 | 77.8 [75.8 to 79.6] | 85.8 [77.7 to 91.9]
  Week 8: number analyzed (Participants) | 1852 | 106
  Week 8 | 80.2 [78.3 to 82.0] | 92.5 [85.7 to 96.7]
  Week 12: number analyzed (Participants) | 1829 | 109
  Week 12 | 80.3 [78.4 to 82.1] | 91.7 [84.9 to 96.2]
  Week 24: number analyzed (Participants) | 1787 | 109
  Week 24 | 82.9 [81.1 to 84.6] | 88.1 [80.5 to 93.5]
  Week 36: number analyzed (Participants) | 1730 | 109
  Week 36 | 82.8 [80.9 to 84.5] | 91.7 [84.9 to 96.2]
  Week 48: number analyzed (Participants) | 1670 | 107
  Week 48 | 82.9 [81.0 to 84.7] | 85.0 [76.9 to 91.2]
  Week 60: number analyzed (Participants) | 1618 | 103
  Week 60 | 84.6 [82.8 to 86.3] | 93.2 [86.5 to 97.2]
  Week 72: number analyzed (Participants) | 1586 | 101
  Week 72 | 84.4 [82.5 to 86.1] | 94.1 [87.5 to 97.8]
  Week 84: number analyzed (Participants) | 1550 | 95
  Week 84 | 84.5 [82.6 to 86.2] | 94.7 [88.1 to 98.3]
  Week 96: number analyzed (Participants) | 1510 | 92
  Week 96 | 85.2 [83.3 to 87.0] | 91.3 [83.6 to 96.2]
  Week 120: number analyzed (Participants) | 1456 | 88
  Week 120 | 84.9 [82.9 to 86.7] | 90.9 [82.9 to 96.0]
  Week 144: number analyzed (Participants) | 1389 | 83
  Week 144 | 86.4 [84.5 to 88.2] | 94.0 [86.5 to 98.0]
  Week 168: number analyzed (Participants) | 1322 | 81
  Week 168 | 86.0 [84.0 to 87.8] | 90.1 [81.5 to 95.6]
  Week 192: number analyzed (Participants) | 1263 | 75
  Week 192 | 85.7 [83.7 to 87.6] | 89.3 [80.1 to 95.3]
  Week 216: number analyzed (Participants) | 1189 | 74
  Week 216 | 87.1 [85.1 to 89.0] | 89.2 [79.8 to 95.2]
  Week 240: number analyzed (Participants) | 1125 | 74
  Week 240 | 86.4 [84.3 to 88.4] | 91.9 [83.2 to 97.0]
  Week 264: number analyzed (Participants) | 1049 | 61
  Week 264 | 88.5 [86.4 to 90.3] | 90.2 [79.8 to 96.3]

7. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50 (ACR50) Response
Description: ACR50 response: >=50% improvement in both TJC and SJC, and >=50% improvement in at least 3 of the 5 remaining ACR core measures assessments: CRP level (in mg/L); participant's assessment of pain (measured on 0 [no pain] to 100 mm [worst pain] VAS); participant's global assessment of disease activity (measured on 0 [no arthritis activity] to 100 mm [maximal arthritis activity] VAS); physician's global assessment of disease activity (measured on 0 [no arthritis activity] to 100 mm [maximal arthritis activity] VAS); participant's assessment of physical function (measured by HAQ-DI, with scoring range of 0 [better physical function] to 3 [worst physical function]). Higher score indicated worse outcomes.
Time Frame: At Week 0 (post-dose), 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240 and 264 of LTS11210
Population: Analysis was performed on safety population. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure and 'number analyzed' = participants with available data for each specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sarilumab + Disease Modifying Anti-Rheumatic Drugs (DMARD) | Sarilumab Monotherapy
Number analyzed (Participants) | 1897 | 111
percentage of participants
  Week 0 | 43.4 [41.2 to 45.7] | 58.6 [48.8 to 67.8]
  Week 4: number analyzed (Participants) | 1884 | 108
  Week 4 | 51.3 [49.0 to 53.6] | 59.3 [49.4 to 68.6]
  Week 8: number analyzed (Participants) | 1850 | 105
  Week 8 | 55.1 [52.8 to 57.4] | 59.0 [49.0 to 68.5]
  Week 12: number analyzed (Participants) | 1830 | 108
  Week 12 | 58.1 [55.8 to 60.4] | 66.7 [56.9 to 75.4]
  Week 24: number analyzed (Participants) | 1782 | 109
  Week 24 | 60.5 [58.2 to 62.8] | 64.2 [54.5 to 73.2]
  Week 36: number analyzed (Participants) | 1729 | 109
  Week 36 | 62.1 [59.8 to 64.4] | 64.2 [54.5 to 73.2]
  Week 48: number analyzed (Participants) | 1669 | 107
  Week 48 | 62.4 [60.0 to 64.7] | 69.2 [59.5 to 77.7]
  Week 60: number analyzed (Participants) | 1620 | 103
  Week 60 | 63.2 [60.8 to 65.6] | 68.9 [59.1 to 77.7]
  Week 72: number analyzed (Participants) | 1585 | 101
  Week 72 | 64.8 [62.4 to 67.1] | 71.3 [61.4 to 79.9]
  Week 84: number analyzed (Participants) | 1546 | 94
  Week 84 | 63.6 [61.2 to 66.1] | 73.4 [63.3 to 82.0]
  Week 96: number analyzed (Participants) | 1511 | 92
  Week 96 | 65.3 [62.8 to 67.7] | 71.7 [61.4 to 80.6]
  Week 120: number analyzed (Participants) | 1455 | 87
  Week 120 | 65.6 [63.1 to 68.0] | 73.6 [63.0 to 82.4]
  Week 144: number analyzed (Participants) | 1385 | 84
  Week 144 | 65.7 [63.1 to 68.2] | 70.2 [59.3 to 79.7]
  Week 168: number analyzed (Participants) | 1320 | 80
  Week 168 | 66.2 [63.6 to 68.8] | 70.0 [58.7 to 79.7]
  Week 192: number analyzed (Participants) | 1257 | 75
  Week 192 | 68.4 [65.8 to 71.0] | 70.7 [59.0 to 80.6]
  Week 216: number analyzed (Participants) | 1189 | 74
  Week 216 | 69.0 [66.3 to 71.7] | 75.7 [64.3 to 84.9]
  Week 240: number analyzed (Participants) | 1125 | 74
  Week 240 | 68.3 [65.5 to 71.0] | 79.7 [68.8 to 88.2]
  Week 264: number analyzed (Participants) | 1040 | 60
  Week 264 | 69.6 [66.7 to 72.4] | 71.7 [58.6 to 82.5]

8. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70 (ACR70) Response
Description: ACR70 response: >=70% improvement in both TJC and SJC, and >=70% improvement in at least 3 of the 5 remaining ACR core measures assessments: CRP level (in mg/L); participant's assessment of pain (measured on 0 [no pain] to 100 mm [worst pain] VAS); participant's global assessment of disease activity (measured on 0 [no arthritis activity]to 100 mm [maximal arthritis activity] VAS); physician's global assessment of disease activity (measured on 0 [no arthritis activity] to 100 mm [maximal arthritis activity] VAS); participant's assessment of physical function (measured by HAQ-DI, with scoring range of 0 [better physical function] to 3 [worst physical function]). Higher score indicated worse outcomes.
Time Frame: At Week 0 (post-dose), 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240 and 264 of LTS11210
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sarilumab + Disease Modifying Anti-Rheumatic Drugs (DMARD) | Sarilumab Monotherapy
Number analyzed (Participants) | 1901 | 111
percentage of participants
  Week 0 | 22.9 [21.0 to 24.8] | 32.4 [23.9 to 42.0]
  Week 4: number analyzed (Participants) | 1879 | 108
  Week 4 | 27.8 [25.8 to 29.9] | 31.5 [22.9 to 41.1]
  Week 8: number analyzed (Participants) | 1854 | 105
  Week 8 | 32.1 [30.0 to 34.3] | 36.2 [27.0 to 46.1]
  Week 12: number analyzed (Participants) | 1829 | 107
  Week 12 | 34.1 [31.9 to 36.3] | 43.0 [33.5 to 52.9]
  Week 24: number analyzed (Participants) | 1781 | 107
  Week 24 | 38.7 [36.4 to 41.0] | 37.4 [28.2 to 47.3]
  Week 36: number analyzed (Participants) | 1726 | 109
  Week 36 | 40.2 [37.9 to 42.6] | 40.4 [31.1 to 50.2]
  Week 48: number analyzed (Participants) | 1666 | 105
  Week 48 | 40.6 [38.3 to 43.0] | 43.8 [34.1 to 53.8]
  Week 60: number analyzed (Participants) | 1618 | 103
  Week 60 | 41.6 [39.2 to 44.0] | 45.6 [35.8 to 55.7]
  Week 72: number analyzed (Participants) | 1585 | 100
  Week 72 | 42.1 [39.6 to 44.6] | 49.0 [38.9 to 59.2]
  Week 84: number analyzed (Participants) | 1541 | 94
  Week 84 | 41.8 [39.3 to 44.3] | 52.1 [41.6 to 62.5]
  Week 96: number analyzed (Participants) | 1510 | 92
  Week 96 | 43.4 [40.9 to 45.9] | 55.4 [44.7 to 65.8]
  Week 120: number analyzed (Participants) | 1449 | 88
  Week 120 | 42.9 [40.3 to 45.5] | 56.8 [45.8 to 67.3]
  Week 144: number analyzed (Participants) | 1386 | 84
  Week 144 | 44.7 [42.0 to 47.3] | 50.0 [38.9 to 61.1]
  Week 168: number analyzed (Participants) | 1317 | 80
  Week 168 | 45.6 [42.9 to 48.4] | 51.3 [39.8 to 62.6]
  Week 192: number analyzed (Participants) | 1262 | 76
  Week 192 | 47.9 [45.1 to 50.7] | 53.9 [42.1 to 65.5]
  Week 216: number analyzed (Participants) | 1186 | 71
  Week 216 | 46.8 [43.9 to 49.7] | 62.0 [49.7 to 73.2]
  Week 240: number analyzed (Participants) | 1123 | 74
  Week 240 | 47.9 [44.9 to 50.9] | 60.8 [48.8 to 72.0]
  Week 264: number analyzed (Participants) | 1030 | 60
  Week 264 | 48.8 [45.7 to 51.9] | 58.3 [44.9 to 70.9]

9. Secondary Outcome: Percentage of Participants With Disease Activity Score for 28 Joints (DAS28) Remission
Description: Disease activity score based on 28 joints and C-reactive protein (DAS28-CRP) was a composite score which included 4 components: TJC with 28 joints assessed; SJC with 28 joints assessed; high-sensitivity CRP (in mg/L) and general health assessment by the participant using participant global assessment (measured on 0 [no arthritis activity] to 100 mm [maximal arthritis activity] VAS). DAS28-CRP total score ranges from 0 to 10, where higher scores indicated greater disease activity. Percentage of participants with DAS28 remission were reported.
Time Frame: At Week 0 (post-dose), 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240, 264, 288, 312, 336, 360, 384, 408, 432, 456, 480, 504 and 516 of LTS11210
Population: Analysis was performed on safety population. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure and 'number analyzed' = participants with available data for each specified category and "0" in the number analyzed field denotes that data were not planned to be collected and analyzed for the specified time-points in the respective groups.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sarilumab + Disease Modifying Anti-Rheumatic Drugs (DMARD) | Sarilumab Monotherapy
Number analyzed (Participants) | 1873 | 110
percentage of participants
  Week 0 | 30.4 [28.3 to 32.5] | 46.4 [36.8 to 56.1]
  Week 4: number analyzed (Participants) | 1867 | 106
  Week 4 | 39.2 [36.9 to 41.4] | 51.9 [42.0 to 61.7]
  Week 8: number analyzed (Participants) | 1804 | 105
  Week 8 | 44.6 [42.3 to 46.9] | 49.5 [39.6 to 59.5]
  Week 12: number analyzed (Participants) | 1819 | 109
  Week 12 | 47.9 [45.6 to 50.3] | 55.0 [45.2 to 64.6]
  Week 24: number analyzed (Participants) | 1778 | 109
  Week 24 | 50.6 [48.2 to 52.9] | 59.6 [49.8 to 68.9]
  Week 36: number analyzed (Participants) | 1721 | 109
  Week 36 | 51.7 [49.3 to 54.1] | 59.6 [49.8 to 68.9]
  Week 48: number analyzed (Participants) | 1661 | 107
  Week 48 | 53.7 [51.3 to 56.1] | 56.1 [46.1 to 65.7]
  Week 60: number analyzed (Participants) | 1608 | 102
  Week 60 | 56.5 [54.1 to 59.0] | 61.8 [51.6 to 71.2]
  Week 72: number analyzed (Participants) | 1580 | 101
  Week 72 | 55.8 [53.3 to 58.3] | 68.3 [58.3 to 77.2]
  Week 84: number analyzed (Participants) | 1537 | 95
  Week 84 | 55.8 [53.2 to 58.3] | 70.5 [60.3 to 79.4]
  Week 96: number analyzed (Participants) | 1506 | 92
  Week 96 | 57.0 [54.5 to 59.6] | 71.7 [61.4 to 80.6]
  Week 120: number analyzed (Participants) | 1444 | 88
  Week 120 | 59.2 [56.6 to 61.8] | 73.9 [63.4 to 82.7]
  Week 144: number analyzed (Participants) | 1381 | 83
  Week 144 | 59.3 [56.7 to 61.9] | 72.3 [61.4 to 81.6]
  Week 168: number analyzed (Participants) | 1309 | 81
  Week 168 | 59.7 [56.9 to 62.3] | 70.4 [59.2 to 80.0]
  Week 192: number analyzed (Participants) | 1250 | 76
  Week 192 | 62.1 [59.3 to 64.8] | 67.1 [55.4 to 77.5]
  Week 216: number analyzed (Participants) | 1175 | 73
  Week 216 | 63.6 [60.7 to 66.3] | 71.2 [59.4 to 81.2]
  Week 240: number analyzed (Participants) | 1118 | 73
  Week 240 | 61.6 [58.7 to 64.5] | 82.2 [71.5 to 90.2]
  Week 264: number analyzed (Participants) | 1036 | 62
  Week 264 | 64.4 [61.4 to 67.3] | 75.8 [63.3 to 85.8]
  Week 288: number analyzed (Participants) | 715 | 26
  Week 288 | 68.7 [65.1 to 72.1] | 73.1 [52.2 to 88.4]
  Week 312: number analyzed (Participants) | 655 | 7
  Week 312 | 69.0 [65.3 to 72.5] | 85.7 [42.1 to 99.6]
  Week 336: number analyzed (Participants) | 540 | 0
  Week 336 | 72.2 [68.2 to 76.0] |
  Week 360: number analyzed (Participants) | 424 | 0
  Week 360 | 71.7 [67.2 to 75.9] |
  Week 384: number analyzed (Participants) | 334 | 0
  Week 384 | 71.6 [66.4 to 76.3] |
  Week 408: number analyzed (Participants) | 199 | 0
  Week 408 | 69.8 [63.0 to 76.1] |
  Week 432: number analyzed (Participants) | 106 | 0
  Week 432 | 76.4 [67.2 to 84.1] |
  Week 456: number analyzed (Participants) | 55 | 0
  Week 456 | 72.7 [59.0 to 83.9] |
  Week 480: number analyzed (Participants) | 39 | 0
  Week 480 | 76.9 [60.7 to 88.9] |
  Week 504: number analyzed (Participants) | 26 | 0
  Week 504 | 73.1 [52.2 to 88.4] |
  Week 516: number analyzed (Participants) | 2 | 0
  Week 516 | 50.0 [1.3 to 98.7] |

10. Secondary Outcome: Percentage of Participants Achieving Good Response, Moderate Response or Non-response Using the European League Against Rheumatism (EULAR) Response Criteria
Description: DAS28-based EULAR response criteria were used to measure individual response as none, good or moderate, depending on the extent of change from baseline and level of disease activity reached. The EULAR response criteria are defined as:
  * Good response = change from baseline of >1.2 and a present DAS28-CRP score <=3.2.
  * Moderate response = change from baseline of >0.6 to <=1.2 and a present DAS28-CRP score <=5.1, or, change from baseline of >1.2 and present DAS28-CRP score >3.2.
  * Non-response = change from baseline of <=0.6, or change from baseline of >0.6 to <=1.2 and present DAS28-CRP score >5.1.
  Scores of good and moderate were considered to indicate therapeutic response. DAS28-CRP is a composite score which included 4 components: TJC with 28 joints assessed; SJC with 28 joints assessed; high-sensitivity CRP (in mg/L) and general health assessment by participant using participant global assessment (measured on 0 [no arthritis activity] to 100 mm [maximal arthritis activity] VAS.
Time Frame: as for outcome 9
Population: Analysis was performed on safety population. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure and 'number analyzed' = participants with available data for each specified category and "0" in the number analyzed field denotes that data was not planned to be collected and analyzed for the specified time-points in the respective groups.
Measure: Number; unit: percentage of participants
Arm/Group | Sarilumab + Disease Modifying Anti-Rheumatic Drugs (DMARD) | Sarilumab Monotherapy
Number analyzed (Participants) | 1872 | 110
percentage of participants
  Week 0: Good response | 44.7 | 60.9
  Week 0: Moderate response | 40.3 | 30.9
  Week 0: None response | 15.0 | 8.2
  Week 4: Good response: number analyzed (Participants) | 1866 | 106
  Week 4: Good response | 57.2 | 69.8
  Week 4: Moderate response: number analyzed (Participants) | 1866 | 106
  Week 4: Moderate response | 36.2 | 26.4
  Week 4:None response: number analyzed (Participants) | 1866 | 106
  Week 4:None response | 6.6 | 3.8
  Week 8: Good response: number analyzed (Participants) | 1803 | 105
  Week 8: Good response | 62.3 | 68.6
  Week 8: Moderate response: number analyzed (Participants) | 1803 | 105
  Week 8: Moderate response | 31.7 | 27.6
  Week 8: None response: number analyzed (Participants) | 1803 | 105
  Week 8: None response | 6.0 | 3.8
  Week 12: Good response: number analyzed (Participants) | 1818 | 109
  Week 12: Good response | 64.1 | 74.3
  Week 12: Moderate response: number analyzed (Participants) | 1818 | 109
  Week 12: Moderate response | 30.6 | 22.9
  Week 12: None response: number analyzed (Participants) | 1818 | 109
  Week 12: None response | 5.2 | 2.8
  Week 24: Good response: number analyzed (Participants) | 1777 | 109
  Week 24: Good response | 66.6 | 73.4
  Week 24: Moderate response: number analyzed (Participants) | 1777 | 109
  Week 24: Moderate response | 28.9 | 24.8
  Week 24: None response: number analyzed (Participants) | 1777 | 109
  Week 24: None response | 4.5 | 1.8
  Week 36: Good response: number analyzed (Participants) | 1720 | 109
  Week 36: Good response | 67.9 | 71.6
  Week 36: Moderate response: number analyzed (Participants) | 1720 | 109
  Week 36: Moderate response | 27.0 | 24.8
  Week 36: None response: number analyzed (Participants) | 1720 | 109
  Week 36: None response | 5.1 | 3.7
  Week 48: Good response: number analyzed (Participants) | 1660 | 107
  Week 48: Good response | 68.1 | 72.0
  Week 48: Moderate response: number analyzed (Participants) | 1660 | 107
  Week 48: Moderate response | 27.4 | 24.3
  Week 48: None response: number analyzed (Participants) | 1660 | 107
  Week 48: None response | 4.5 | 3.7
  Week 60: Good response: number analyzed (Participants) | 1607 | 102
  Week 60: Good response | 71.1 | 68.6
  Week 60: Moderate response: number analyzed (Participants) | 1607 | 102
  Week 60: Moderate response | 24.6 | 29.4
  Week 60: None response: number analyzed (Participants) | 1607 | 102
  Week 60: None response | 4.2 | 2.0
  Week 72: Good response: number analyzed (Participants) | 1579 | 101
  Week 72: Good response | 70.0 | 81.2
  Week 72: Moderate response: number analyzed (Participants) | 1579 | 101
  Week 72: Moderate response | 26.0 | 16.8
  Week 72: None response: number analyzed (Participants) | 1579 | 101
  Week 72: None response | 4.0 | 2.0
  Week 84: Good response: number analyzed (Participants) | 1536 | 95
  Week 84: Good response | 71.3 | 84.2
  Week 84: Moderate response: number analyzed (Participants) | 1536 | 95
  Week 84: Moderate response | 24.2 | 14.7
  Week 84: None response: number analyzed (Participants) | 1536 | 95
  Week 84: None response | 4.6 | 1.1
  Week 96: Good response: number analyzed (Participants) | 1505 | 92
  Week 96: Good response | 72.6 | 76.1
  Week 96: Moderate response: number analyzed (Participants) | 1505 | 92
  Week 96: Moderate response | 23.3 | 21.7
  Week 96: None response: number analyzed (Participants) | 1505 | 92
  Week 96: None response | 4.1 | 2.2
  Week 120: Good response: number analyzed (Participants) | 1443 | 88
  Week 120: Good response | 73.5 | 80.7
  Week 120: Moderate response: number analyzed (Participants) | 1443 | 88
  Week 120: Moderate response | 22.3 | 17.0
  Week 120: None response: number analyzed (Participants) | 1443 | 88
  Week 120: None response | 4.2 | 2.3
  Week 144: Good response: number analyzed (Participants) | 1381 | 83
  Week 144: Good response | 73.3 | 86.7
  Week 144: Moderate response: number analyzed (Participants) | 1381 | 83
  Week 144: Moderate response | 22.8 | 13.3
  Week 144: None response: number analyzed (Participants) | 1381 | 83
  Week 144: None response | 3.9 | 0
  Week 168: Good response: number analyzed (Participants) | 1309 | 81
  Week 168: Good response | 74.5 | 84.0
  Week 168: Moderate response: number analyzed (Participants) | 1309 | 81
  Week 168: Moderate response | 20.6 | 16.0
  Week 168: None response: number analyzed (Participants) | 1309 | 81
  Week 168: None response | 4.9 | 0
  Week 192: Good response: number analyzed (Participants) | 1250 | 76
  Week 192: Good response | 75.6 | 81.6
  Week 192: Moderate response: number analyzed (Participants) | 1250 | 76
  Week 192: Moderate response | 20.6 | 13.2
  Week 192: None response: number analyzed (Participants) | 1250 | 76
  Week 192: None response | 3.8 | 5.3
  Week 216: Good response: number analyzed (Participants) | 1175 | 73
  Week 216: Good response | 75.9 | 80.8
  Week 216: Moderate response: number analyzed (Participants) | 1175 | 73
  Week 216: Moderate response | 20.5 | 17.8
  Week 216: None response: number analyzed (Participants) | 1175 | 73
  Week 216: None response | 3.6 | 1.4
  Week 240: Good response: number analyzed (Participants) | 1118 | 73
  Week 240: Good response | 78.6 | 89.0
  Week 240: Moderate response: number analyzed (Participants) | 1118 | 73
  Week 240: Moderate response | 17.5 | 9.6
  Week 240: None response: number analyzed (Participants) | 1118 | 73
  Week 240: None response | 3.8 | 1.4
  Week 264: Good response: number analyzed (Participants) | 1036 | 62
  Week 264: Good response | 76.7 | 83.9
  Week 264: Moderate response: number analyzed (Participants) | 1036 | 62
  Week 264: Moderate response | 20.2 | 16.1
  Week 264: None response: number analyzed (Participants) | 1036 | 62
  Week 264: None response | 3.1 | 0
  Week 288: Good response: number analyzed (Participants) | 715 | 26
  Week 288: Good response | 82.4 | 80.8
  Week 288: Moderate response: number analyzed (Participants) | 715 | 26
  Week 288: Moderate response | 15.2 | 19.2
  Week 288: None response: number analyzed (Participants) | 715 | 26
  Week 288: None response | 2.4 | 0
  Week 312: Good response: number analyzed (Participants) | 655 | 7
  Week 312: Good response | 81.5 | 100
  Week 312: Moderate response: number analyzed (Participants) | 655 | 7
  Week 312: Moderate response | 16.3 | 0
  Week 312: None response: number analyzed (Participants) | 655 | 7
  Week 312: None response | 2.1 | 0
  Week 336: Good response: number analyzed (Participants) | 540 | 0
  Week 336: Good response | 83.0 |
  Week 336: Moderate response: number analyzed (Participants) | 540 | 0
  Week 336: Moderate response | 14.6 |
  Week 336: None response: number analyzed (Participants) | 540 | 0
  Week 336: None response | 2.4 |
  Week 360: Good response: number analyzed (Participants) | 424 | 0
  Week 360: Good response | 83.3 |
  Week 360: Moderate response: number analyzed (Participants) | 424 | 0
  Week 360: Moderate response | 15.1 |
  Week 360: None response: number analyzed (Participants) | 424 | 0
  Week 360: None response | 1.7 |
  Week 384: Good response: number analyzed (Participants) | 334 | 0
  Week 384: Good response | 86.2 |
  Week 384: Moderate response: number analyzed (Participants) | 334 | 0
  Week 384: Moderate response | 12.9 |
  Week 384: None response: number analyzed (Participants) | 334 | 0
  Week 384: None response | 0.9 |
  Week 408: Good response: number analyzed (Participants) | 199 | 0
  Week 408: Good response | 81.9 |
  Week 408: Moderate response: number analyzed (Participants) | 199 | 0
  Week 408: Moderate response | 16.1 |
  Week 408: None response: number analyzed (Participants) | 199 | 0
  Week 408: None response | 2.0 |
  Week 432: Good response: number analyzed (Participants) | 106 | 0
  Week 432: Good response | 85.8 |
  Week 432: Moderate response: number analyzed (Participants) | 106 | 0
  Week 432: Moderate response | 14.2 |
  Week 432: None response: number analyzed (Participants) | 106 | 0
  Week 432: None response | 0 |
  Week 456: Good response: number analyzed (Participants) | 55 | 0
  Week 456: Good response | 87.3 |
  Week 456: Moderate response: number analyzed (Participants) | 55 | 0
  Week 456: Moderate response | 12.7 |
  Week 456: None response: number analyzed (Participants) | 55 | 0
  Week 456: None response | 0 |
  Week 480: Good response: number analyzed (Participants) | 39 | 0
  Week 480: Good response | 79.5 |
  Week 480: Moderate response: number analyzed (Participants) | 39 | 0
  Week 480: Moderate response | 17.9 |
  Week 480: None response: number analyzed (Participants) | 39 | 0
  Week 480: None response | 2.6 |
  Week 504: Good response: number analyzed (Participants) | 26 | 0
  Week 504: Good response | 92.3 |
  Week 504: Moderate response: number analyzed (Participants) | 26 | 0
  Week 504: Moderate response | 7.7 |
  Week 504: None response: number analyzed (Participants) | 26 | 0
  Week 504: None response | 0 |
  Week 516: Good response: number analyzed (Participants) | 2 | 0
  Week 516: Good response | 100 |
  Week 516: Moderate response: number analyzed (Participants) | 2 | 0
  Week 516: Moderate response | 0 |
  Week 516: None response: number analyzed (Participants) | 2 | 0
  Week 516: None response | 0 |

11. Secondary Outcome: Change From Baseline in DAS28-CRP Score at Weeks 0, 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240, 264, 288, 312, 336, 360, 384, 408, 432, 456, 480, 504 and 516 of LTS11210
Description: DAS28-CRP is a composite score which included 4 components: TJC with 28 joints assessed; SJC with 28 joints assessed; high-sensitivity CRP (in mg/L) and general health assessment by the participant using participant global assessment (measured on 0 [no arthritis activity] to 100 mm [maximal arthritis activity] VAS). DAS28-CRP total score ranges from 0-10, where higher scores indicated greater disease activity. Here, Baseline refers to the Baseline of initial studies (EFC11072, ACT11575, EFC10832, SFY13370 and EFC13752).
Time Frame: Baseline, Week 0 (post-dose), 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240, 264, 288, 312, 336, 360, 384, 408, 432, 456, 480, 504 and 516 of LTS11210
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sarilumab + Disease Modifying Anti-Rheumatic Drugs (DMARD) | Sarilumab Monotherapy
Number analyzed (Participants) | 1872 | 110
units on a scale
  Week 0 | -2.50 (1.52) | -2.99 (1.42)
  Week 4: number analyzed (Participants) | 1866 | 106
  Week 4 | -2.98 (1.38) | -3.18 (1.31)
  Week 8: number analyzed (Participants) | 1803 | 105
  Week 8 | -3.12 (1.41) | -3.21 (1.26)
  Week 12: number analyzed (Participants) | 1818 | 109
  Week 12 | -3.19 (1.41) | -3.28 (1.29)
  Week 24: number analyzed (Participants) | 1777 | 109
  Week 24 | -3.28 (1.41) | -3.43 (1.21)
  Week 36: number analyzed (Participants) | 1720 | 109
  Week 36 | -3.31 (1.43) | -3.35 (1.23)
  Week 48: number analyzed (Participants) | 1660 | 107
  Week 48 | -3.35 (1.42) | -3.36 (1.35)
  Week 60: number analyzed (Participants) | 1607 | 102
  Week 60 | -3.41 (1.41) | -3.50 (1.28)
  Week 72: number analyzed (Participants) | 1579 | 101
  Week 72 | -3.41 (1.42) | -3.61 (1.24)
  Week 84: number analyzed (Participants) | 1536 | 95
  Week 84 | -3.40 (1.45) | -3.70 (1.19)
  Week 96: number analyzed (Participants) | 1505 | 92
  Week 96 | -3.46 (1.43) | -3.59 (1.32)
  Week 120: number analyzed (Participants) | 1443 | 88
  Week 120 | -3.49 (1.45) | -3.72 (1.20)
  Week 144: number analyzed (Participants) | 1381 | 83
  Week 144 | -3.51 (1.41) | -3.79 (1.29)
  Week 168: number analyzed (Participants) | 1309 | 81
  Week 168 | -3.52 (1.45) | -3.66 (1.30)
  Week 192: number analyzed (Participants) | 1250 | 76
  Week 192 | -3.55 (1.43) | -3.61 (1.48)
  Week 216: number analyzed (Participants) | 1175 | 73
  Week 216 | -3.59 (1.43) | -3.71 (1.24)
  Week 240: number analyzed (Participants) | 1118 | 73
  Week 240 | -3.57 (1.44) | -3.90 (1.35)
  Week 264: number analyzed (Participants) | 1036 | 62
  Week 264 | -3.64 (1.39) | -3.92 (1.36)
  Week 288: number analyzed (Participants) | 715 | 26
  Week 288 | -3.80 (1.38) | -4.38 (1.33)
  Week 312: number analyzed (Participants) | 655 | 7
  Week 312 | -3.86 (1.34) | -5.62 (0.86)
  Week 336: number analyzed (Participants) | 540 | 0
  Week 336 | -3.86 (1.34) |
  Week 360: number analyzed (Participants) | 424 | 0
  Week 360 | -3.93 (1.34) |
  Week 384: number analyzed (Participants) | 334 | 0
  Week 384 | -3.99 (1.36) |
  Week 408: number analyzed (Participants) | 199 | 0
  Week 408 | -3.85 (1.44) |
  Week 432: number analyzed (Participants) | 106 | 0
  Week 432 | -4.11 (1.35) |
  Week 456: number analyzed (Participants) | 55 | 0
  Week 456 | -4.01 (1.14) |
  Week 480: number analyzed (Participants) | 39 | 0
  Week 480 | -3.69 (1.47) |
  Week 504: number analyzed (Participants) | 26 | 0
  Week 504 | -3.76 (1.24) |
  Week 516: number analyzed (Participants) | 2 | 0
  Week 516 | -3.76 (2.32) |

12. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Scores at Week 0, 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240 and 264 of LTS11210
Description: HAQ-DI is a standardized questionnaire used to assess the degree of difficulty a participant has experienced during the past week in 8 domains of daily living activities: dressing/grooming; arising; eating; walking; hygiene; reach; grip and activities. There were total of 30 items distributed in these 8 domains. Each item was scored on a 4-point scale from 0 to 3, where 0= no difficulty in physical function; 1= some difficulty in physical function; 2= much difficulty in physical function; 3= unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0 (least difficulty in physical function) to 3 (extreme difficulty in physical function), where higher scores indicate more difficulty while performing daily living activities. Here, Baseline refers to the Baseline of initial studies (EFC11072, ACT11575, EFC10832, SFY13370 and EFC13752).
Time Frame: Baseline, Week 0 (post-dose), 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240 and 264 of LTS11210
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sarilumab + Disease Modifying Anti-Rheumatic Drugs (DMARD) | Sarilumab Monotherapy
Number analyzed (Participants) | 1895 | 111
units on a scale
  Week 0 | -0.56 (0.63) | -0.58 (0.59)
  Week 4: number analyzed (Participants) | 1882 | 109
  Week 4 | -0.59 (0.62) | -0.57 (0.52)
  Week 8: number analyzed (Participants) | 1858 | 106
  Week 8 | -0.63 (0.63) | -0.63 (0.53)
  Week 12: number analyzed (Participants) | 1826 | 109
  Week 12 | -0.65 (0.64) | -0.65 (0.57)
  Week 24: number analyzed (Participants) | 1787 | 109
  Week 24 | -0.69 (0.65) | -0.63 (0.60)
  Week 36: number analyzed (Participants) | 1728 | 109
  Week 36 | -0.70 (0.66) | -0.67 (0.61)
  Week 48: number analyzed (Participants) | 1667 | 107
  Week 48 | -0.70 (0.66) | -0.63 (0.60)
  Week 60: number analyzed (Participants) | 1625 | 103
  Week 60 | -0.70 (0.67) | -0.67 (0.50)
  Week 72: number analyzed (Participants) | 1586 | 101
  Week 72 | -0.71 (0.66) | -0.67 (0.59)
  Week 84: number analyzed (Participants) | 1551 | 95
  Week 84 | -0.71 (0.68) | -0.68 (0.59)
  Week 96: number analyzed (Participants) | 1509 | 92
  Week 96 | -0.72 (0.67) | -0.69 (0.58)
  Week 120: number analyzed (Participants) | 1458 | 89
  Week 120 | -0.74 (0.69) | -0.67 (0.55)
  Week 144: number analyzed (Participants) | 1386 | 84
  Week 144 | -0.73 (0.70) | -0.64 (0.61)
  Week 168: number analyzed (Participants) | 1327 | 81
  Week 168 | -0.74 (0.70) | -0.61 (0.59)
  Week 192: number analyzed (Participants) | 1268 | 77
  Week 192 | -0.74 (0.71) | -0.65 (0.65)
  Week 216: number analyzed (Participants) | 1185 | 70
  Week 216 | -0.75 (0.71) | -0.62 (0.69)
  Week 240: number analyzed (Participants) | 1127 | 74
  Week 240 | -0.74 (0.72) | -0.61 (0.64)
  Week 264: number analyzed (Participants) | 998 | 57
  Week 264 | -0.76 (0.71) | -0.54 (0.62)

13. Secondary Outcome: Change From Baseline in Van Der Heijde Modified Total Sharp Score (mTSS) at Week 0 and Week 48 of LTS11210: Campaign 1 X-ray Data - Participants From EFC11072 Part B
Description: Van der Heijde modified Sharp method is composite X-ray scoring system used to assess structural (joint) disease progression in RA. The method evaluates both joint erosions (JE) for 44 joints and joint space narrowing (JSN) for 42 joints in bilateral hand and foot joints. Total mTSS: sum of the scores from both erosion score and joint space narrowing score and ranged from 0 (normal, no progression) to 448 (worst possible total score). An increase in total score represents progression of structural damage. Here, Baseline refers to the Baseline of initial study (EFC11072 Part B). In this outcome measure, change from initial study Baseline in 2 years X-ray data at Week 0 and 48 of LTS11210 were reported.
Time Frame: Baseline, Week 0 and 48 of LTS11210
Population: Analyzed on subset of participants who previously completed study EFC11072, Part B with end of treatment X-ray evaluation. Here, 'overall number of participants analyzed' = participants from studies EFC11072 Part B evaluable for this outcome measure and 'number analyzed' = participants with available data for each specified category. Data for this outcome measure was not planned to be collected and analyzed for Sarilumab Monotherapy arm, as pre-specified in protocol.
Measure: Mean (Standard Deviation); unit: score on scale
Groups:
- Sarilumab + DMARD: EFC11072 Part B: Participants who completed EFC11072 Part B were enrolled in LTS11210 and received sarilumab 150 mg SC qw. Dose could be reduced to 150 mg q2w due to neutropenia, thrombocytopenia or increase in liver enzymes (ALT). After dose regimens selection for Phase 3 studies (150 mg q2w and 200 mg q2w), participants already receiving 150 mg qw were switched to sarilumab 200 mg q2w. Treatment duration per participant was at least 264 weeks from first study drug administration in LTS11210. Participants continued to be treated beyond 264 weeks until sarilumab was commercially available in their respective countries or until 2020, at the latest (maximum duration: 523 weeks). Participants who were already taking concomitant non-biologic DMARDs in initial study continued stable dose of one or combination of conventional synthetic DMARDs they were taking.
Arm/Group | Sarilumab + DMARD: EFC11072 Part B
Number analyzed (Participants) | 856
score on scale
  Change at Week 0 | 1.05 (4.61)
  Change at Week 48: number analyzed (Participants) | 848
  Change at Week 48 | 1.34 (5.31)

14. Secondary Outcome: Change From Baseline in Van Der Heijde Modified Total Sharp Score (mTSS) at Week 48 and Week 96 of LTS11210: Campaign 2 X-ray Data - Participants From EFC11072 Part B
Description: Van der Heijde modified Sharp method is composite X-ray scoring system used to assess structural (joint) disease progression in RA. The method evaluates both JE for 44 joints and JSN for 42 joints in bilateral hand and foot joints. Total mTSS: sum of the scores from both erosion score and joint space narrowing score and ranged from 0 (normal, no progression) to 448 (worst possible total score). An increase in total score represents progression of structural damage. Here, Baseline refers to the Baseline of initial study (EFC11072 Part B). In this outcome measure, change from initial study (EFC11072 Part B) Baseline in 3 years X-ray data (participants with study duration of more than 48 weeks in LTS11210) at Week 48 and 96 of LTS11210 from Campaign 2 were reported.
Time Frame: Baseline, Week 48 and 96 of LTS11210
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Sarilumab + DMARD: EFC11072 Part B
Number analyzed (Participants) | 756
score on scale
  Change at Week 48 | 1.60 (5.96)
  Change at Week 96: number analyzed (Participants) | 755
  Change at Week 96 | 2.14 (7.20)

15. Secondary Outcome: Change From Baseline in Van Der Heijde Modified Total Sharp Score (mTSS) at Week 96, Week 144 and Week 192 of LTS11210: Campaign 3 X-ray Data - Participants From EFC11072 Part B
Description: Van der Heijde modified Sharp method is composite X-ray scoring system used to assess structural (joint) disease progression in RA. The method evaluates both JE for 44 joints and JSN for 42 joints in bilateral hand and foot joints. Total mTSS: sum of the scores from both erosion score and joint space narrowing score and ranged from 0 (normal, no progression) to 448 (worst possible total score). An increase in total score represents progression of structural damage. Here, Baseline refers to the Baseline of initial study (EFC11072 Part B). In this outcome measure, change from initial study (EFC11072 Part B) Baseline in 5 years X-ray data (participants with study duration of more than 96 weeks in LTS11210) at Week 96, 144 and 192 of LTS11210 from Campaign 3 were reported.
Time Frame: Baseline, Week 96, 144 and 192 of LTS11210
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Sarilumab + DMARD: EFC11072 Part B
Number analyzed (Participants) | 699
score on scale
  Change at Week 96 | 1.83 (7.76)
  Change at Week 144: number analyzed (Participants) | 689
  Change at Week 144 | 2.24 (8.43)
  Change at Week 192: number analyzed (Participants) | 656
  Change at Week 192 | 2.83 (9.42)

16. Secondary Outcome: Percentage of Participants With no Radiographic Progression of the Van Der Heijde Modified Total Sharp Score at Week 0 and 48 of LTS11210: Campaign 1 X-ray Data - Participants From EFC11072 Part B
Description: Radiographic no progression: defined as a change from Baseline in Van der Heijde mTSS <= 0. Van der Heijde modified Sharp method is composite X-ray scoring system used to assess structural (joint) disease progression in RA. The method evaluates both JE for 44 joints and JSN for 42 joints in bilateral hand and foot joints. Total mTSS was sum of scores from both erosion score and joint space narrowing score, ranged from 0 (normal, no progression) to 448 (worst possible total score). Increase in total score represents progression of structural damage. In this outcome measure, percentage of participants with no radiographic progression at Week 48 of LTS11210 from Campaign 1 X-ray data were reported.
Time Frame: Week 0 (post-dose) and 48 of LTS11210
Population: Analyzed on subset of participants who previously completed study EFC11072, Part B with end of treatment X-ray evaluation. Here, 'overall number of participants analyzed' = participants from studies EFC11072 Part B evaluable for this outcome measure. Data for this outcome measure was not planned to be collected and analyzed for Sarilumab Monotherapy arm, as pre-specified in protocol.
Measure: Number; unit: percentage of participants
Arm/Group | Sarilumab + DMARD: EFC11072 Part B
Number analyzed (Participants) | 889
percentage of participants
  Week 0 | 51.9
  Week 48 | 51.2

17. Secondary Outcome: Percentage of Participants With no Radiographic Progression of the Van Der Heijde Modified Total Sharp Score at Week 48 and Week 96 of LTS11210: Campaign 2 X-ray Data - Participants From EFC11072 Part B
Description: Radiographic no progression: defined as a change from Baseline in Van der Heijde mTSS <= 0. Van der Heijde modified Sharp method is composite X-ray scoring system used to assess structural (joint) disease progression in RA. The method evaluates both JE for 44 joints and JSN for 42 joints in bilateral hand and foot joints. Total mTSS was sum of scores from both erosion score and joint space narrowing score, ranged from 0 (normal, no progression) to 448 (worst possible total score). Increase in total score represents progression of structural damage. In this outcome measure, percentage of participants with no radiographic progression at Week 48 and 96 of LTS11210 from Campaign 2 X-ray data (participants with study duration of more than 48 weeks in LTS11210) were reported.
Time Frame: Week 48 and 96 of LTS11210
Population: as for outcome 16
Measure: Number; unit: percentage of participants
Arm/Group | Sarilumab + DMARD: EFC11072 Part B
Number analyzed (Participants) | 796
percentage of participants
  Week 48 | 46.6
  Week 96 | 44.2

18. Secondary Outcome: Percentage of Participants With no Radiographic Progression of the Van Der Heijde Modified Total Sharp Score at Week 96, 144 and 192 of LTS11210: Campaign 3 X-ray Data - Participants From EFC11072 Part B
Description: Radiographic no progression: defined as a change from Baseline in Van der Heijde mTSS <= 0. Van der Heijde modified Sharp method is composite X-ray scoring system used to assess structural (joint) disease progression in RA. The method evaluates both JE for 44 joints and JSN for 42 joints in bilateral hand and foot joints. Total mTSS was sum of scores from both erosion score and joint space narrowing score, ranged from 0 (normal, no progression) to 448 (worst possible total score). Increase in total score represents progression of structural damage. In this outcome measure, percentage of participants with no radiographic progression at Week 96, 144 and 192 of LTS11210 from Campaign 3 X-ray data (participants with study duration more than 96 weeks in LTS11210) were reported.
Time Frame: Week 96, 144 and 192 of LTS11210
Population: as for outcome 16
Measure: Number; unit: percentage of participants
Arm/Group | Sarilumab + DMARD: EFC11072 Part B
Number analyzed (Participants) | 732
percentage of participants
  Week 96 | 48.6
  Week 144 | 46.0
  Week 192 | 41.8

19. Secondary Outcome: Change From Baseline in Tender Joint Count (TJC) at Week 0, 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240, 264, 288, 312, 336, 360, 384, 408, 432, 456, 480, 504 and 516 of LTS11210
Description: TJC is the sum of all tender joints based on examination of the 68 joints of the fingers, elbows, hips, knees, ankles, and toes. Total TJC ranged from 0 (best) to 68 (worst), where higher score = more severity. Change from Baseline in TJC was reported in the outcome measure. Here, Baseline refers to Baseline of initial study (EFC11072, ACT11575, EFC10832, SFY13370 and EFC13752).
Time Frame: as for outcome 11
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Sarilumab + Disease Modifying Anti-Rheumatic Drugs (DMARD) | Sarilumab Monotherapy
Number analyzed (Participants) | 1904 | 111
joints
  Week 0 | -16.67 (14.05) | -19.86 (12.43)
  Week 4: number analyzed (Participants) | 1891 | 109
  Week 4 | -18.97 (13.81) | -20.13 (12.64)
  Week 8: number analyzed (Participants) | 1867 | 106
  Week 8 | -19.72 (13.61) | -20.09 (11.73)
  Week 12: number analyzed (Participants) | 1837 | 109
  Week 12 | -20.20 (13.89) | -20.05 (12.99)
  Week 24: number analyzed (Participants) | 1791 | 109
  Week 24 | -20.67 (14.09) | -21.19 (12.55)
  Week 36: number analyzed (Participants) | 1733 | 109
  Week 36 | -20.68 (14.39) | -20.60 (12.19)
  Week 48: number analyzed (Participants) | 1674 | 107
  Week 48 | -20.95 (14.04) | -20.27 (13.54)
  Week 60: number analyzed (Participants) | 1625 | 103
  Week 60 | -21.29 (14.06) | -20.95 (12.66)
  Week 72: number analyzed (Participants) | 1589 | 101
  Week 72 | -21.41 (13.98) | -21.67 (12.65)
  Week 84: number analyzed (Participants) | 1553 | 95
  Week 84 | -21.53 (14.17) | -21.36 (13.04)
  Week 96: number analyzed (Participants) | 1514 | 92
  Week 96 | -21.65 (14.08) | -20.89 (13.50)
  Week 120: number analyzed (Participants) | 1459 | 88
  Week 120 | -21.92 (14.20) | -20.18 (12.73)
  Week 144: number analyzed (Participants) | 1394 | 83
  Week 144 | -22.13 (14.01) | -22.52 (13.41)
  Week 168: number analyzed (Participants) | 1331 | 81
  Week 168 | -22.35 (14.26) | -22.42 (13.34)
  Week 192: number analyzed (Participants) | 1269 | 78
  Week 192 | -22.62 (14.20) | -21.83 (13.79)
  Week 216: number analyzed (Participants) | 1211 | 76
  Week 216 | -22.69 (14.28) | -22.33 (13.29)
  Week 240: number analyzed (Participants) | 1136 | 74
  Week 240 | -22.89 (14.47) | -23.07 (14.24)
  Week 264: number analyzed (Participants) | 1072 | 62
  Week 264 | -23.09 (14.08) | -23.66 (15.02)
  Week 288: number analyzed (Participants) | 788 | 26
  Week 288 | -22.59 (15.70) | -28.95 (14.79)
  Week 312: number analyzed (Participants) | 713 | 7
  Week 312 | -23.47 (15.23) | -43.71 (12.12)
  Week 336: number analyzed (Participants) | 556 | 0
  Week 336 | -23.37 (15.24) |
  Week 360: number analyzed (Participants) | 442 | 0
  Week 360 | -24.12 (14.89) |
  Week 384: number analyzed (Participants) | 358 | 0
  Week 384 | -24.73 (15.14) |
  Week 408: number analyzed (Participants) | 226 | 0
  Week 408 | -24.58 (14.97) |
  Week 432: number analyzed (Participants) | 109 | 0
  Week 432 | -25.33 (15.05) |
  Week 456: number analyzed (Participants) | 59 | 0
  Week 456 | -24.21 (14.37) |
  Week 480: number analyzed (Participants) | 45 | 0
  Week 480 | -21.23 (14.66) |
  Week 504: number analyzed (Participants) | 27 | 0
  Week 504 | -23.62 (13.63) |
  Week 516: number analyzed (Participants) | 2 | 0
  Week 516 | -24.00 (12.73) |

20. Secondary Outcome: Change From Baseline in Swollen Joint Count (SJC) at Week 0, 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240, 264, 288, 312, 336, 360, 384, 408, 432, 456, 480, 504 and 516 of LTS11210
Description: SJC is the sum of all swollen joints based on examination of the fingers, elbows, knees and toes. Total SJC ranged from 0 (best) to 66 (worst), where higher score = more severity. Change from Baseline in SJC was reported in the outcome measure. Here, Baseline refers to the Baseline of initial studies (EFC11072, ACT11575, EFC10832, SFY13370 and EFC13752).
Time Frame: as for outcome 11
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Sarilumab + Disease Modifying Anti-Rheumatic Drugs (DMARD) | Sarilumab Monotherapy
Number analyzed (Participants) | 1904 | 111
joints
  Week 0 | -11.36 (9.96) | -14.06 (9.65)
  Week 4: number analyzed (Participants) | 1891 | 109
  Week 4 | -12.81 (9.77) | -14.55 (9.19)
  Week 8: number analyzed (Participants) | 1867 | 106
  Week 8 | -13.43 (9.82) | -14.60 (9.30)
  Week 12: number analyzed (Participants) | 1837 | 109
  Week 12 | -13.77 (10.13) | -14.58 (9.31)
  Week 24: number analyzed (Participants) | 1791 | 109
  Week 24 | -14.28 (10.09) | -14.83 (9.64)
  Week 36: number analyzed (Participants) | 1733 | 109
  Week 36 | -14.37 (9.99) | -14.51 (9.70)
  Week 48: number analyzed (Participants) | 1674 | 107
  Week 48 | -14.53 (9.97) | -14.96 (9.22)
  Week 60: number analyzed (Participants) | 1625 | 103
  Week 60 | -14.75 (10.20) | -15.54 (9.49)
  Week 72: number analyzed (Participants) | 1589 | 101
  Week 72 | -14.76 (10.12) | -15.43 (9.67)
  Week 84: number analyzed (Participants) | 1553 | 95
  Week 84 | -14.84 (10.16) | -15.83 (9.50)
  Week 96: number analyzed (Participants) | 1514 | 92
  Week 96 | -15.03 (10.20) | -15.51 (10.24)
  Week 120: number analyzed (Participants) | 1459 | 88
  Week 120 | -15.09 (10.17) | -15.77 (9.95)
  Week 144: number analyzed (Participants) | 1394 | 83
  Week 144 | -15.18 (10.20) | -15.90 (8.57)
  Week 168: number analyzed (Participants) | 1331 | 81
  Week 168 | -15.16 (10.30) | -15.47 (8.91)
  Week 192: number analyzed (Participants) | 1269 | 78
  Week 192 | -15.26 (10.09) | -15.01 (9.17)
  Week 216: number analyzed (Participants) | 1211 | 76
  Week 216 | -15.25 (9.97) | -15.72 (8.65)
  Week 240: number analyzed (Participants) | 1135 | 74
  Week 240 | -15.43 (10.34) | -15.59 (9.08)
  Week 264: number analyzed (Participants) | 1072 | 62
  Week 264 | -15.50 (9.79) | -16.59 (9.53)
  Week 288: number analyzed (Participants) | 788 | 26
  Week 288 | -14.67 (10.98) | -18.65 (8.90)
  Week 312: number analyzed (Participants) | 713 | 7
  Week 312 | -15.38 (10.71) | -23.57 (9.83)
  Week 336: number analyzed (Participants) | 556 | 0
  Week 336 | -15.51 (10.48) |
  Week 360: number analyzed (Participants) | 442 | 0
  Week 360 | -15.96 (10.76) |
  Week 384: number analyzed (Participants) | 358 | 0
  Week 384 | -16.42 (10.76) |
  Week 408: number analyzed (Participants) | 226 | 0
  Week 408 | -16.30 (11.47) |
  Week 432: number analyzed (Participants) | 109 | 0
  Week 432 | -16.62 (11.51) |
  Week 456: number analyzed (Participants) | 59 | 0
  Week 456 | -15.64 (10.65) |
  Week 480: number analyzed (Participants) | 45 | 0
  Week 480 | -15.43 (10.67) |
  Week 504: number analyzed (Participants) | 27 | 0
  Week 504 | -16.21 (10.94) |
  Week 516: number analyzed (Participants) | 2 | 0
  Week 516 | -13.00 (2.83) |

21. Secondary Outcome: Change From Baseline in Physician's Global Assessments of Disease Activity Visual Analogue Scale (VAS) Score at Week 0, 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240, and 264 of LTS11210
Description: Physician global assessment of disease activity was measured on a 100 millimeters (mm) horizontal VAS, ranging from 0 (best disease activity) to 100 (worst disease activity), where lower score = less disease activity and higher score = more disease activity. Here, Baseline refers to Baseline of initial studies (EFC11072, ACT11575, EFC10832, SFY13370 and EFC13752).
Time Frame: Baseline, Week 0 (post-dose), 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240, and 264 of LTS11210
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Sarilumab + Disease Modifying Anti-Rheumatic Drugs (DMARD) | Sarilumab Monotherapy
Number analyzed (Participants) | 1903 | 110
millimeters
  Week 0 | -40.51 (23.82) | -46.38 (19.17)
  Week 4: number analyzed (Participants) | 1888 | 109
  Week 4 | -43.98 (22.03) | -47.94 (19.16)
  Week 8: number analyzed (Participants) | 1863 | 106
  Week 8 | -45.79 (22.06) | -49.27 (18.80)
  Week 12: number analyzed (Participants) | 1832 | 109
  Week 12 | -47.02 (22.03) | -50.20 (19.74)
  Week 24: number analyzed (Participants) | 1786 | 109
  Week 24 | -48.39 (21.94) | -50.82 (19.99)
  Week 36: number analyzed (Participants) | 1730 | 109
  Week 36 | -48.94 (21.72) | -51.12 (19.87)
  Week 48: number analyzed (Participants) | 1675 | 107
  Week 48 | -49.36 (21.68) | -50.58 (21.38)
  Week 60: number analyzed (Participants) | 1624 | 103
  Week 60 | -49.98 (21.62) | -51.40 (20.51)
  Week 72: number analyzed (Participants) | 1586 | 101
  Week 72 | -49.91 (21.72) | -52.90 (19.40)
  Week 84: number analyzed (Participants) | 1551 | 94
  Week 84 | -50.28 (21.42) | -55.84 (17.39)
  Week 96: number analyzed (Participants) | 1512 | 92
  Week 96 | -50.73 (21.62) | -54.14 (18.97)
  Week 120: number analyzed (Participants) | 1458 | 88
  Week 120 | -50.43 (21.39) | -54.33 (19.41)
  Week 144: number analyzed (Participants) | 1390 | 84
  Week 144 | -50.84 (21.13) | -55.73 (18.04)
  Week 168: number analyzed (Participants) | 1329 | 81
  Week 168 | -50.49 (21.65) | -53.21 (21.36)
  Week 192: number analyzed (Participants) | 1264 | 78
  Week 192 | -50.32 (22.00) | -52.22 (22.44)
  Week 216: number analyzed (Participants) | 1209 | 76
  Week 216 | -51.49 (21.57) | -54.67 (18.30)
  Week 240: number analyzed (Participants) | 1133 | 74
  Week 240 | -51.00 (21.57) | -55.16 (18.82)
  Week 264: number analyzed (Participants) | 1055 | 63
  Week 264 | -51.18 (21.24) | -55.27 (21.70)

22. Secondary Outcome: Change From Baseline in Participant Global Assessment of Disease Activity Visual Analogue Scale Score at Week 0, 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240, 264, 288, 312, 336, 360, 384, 408, 432, 456, 480, 504 and 516 of LTS11210
Description: Participant global assessment of disease activity was measured on a 100 mm horizontal VAS, ranging from 0 (best disease activity) to 100 (worst disease activity), where lower score = less disease activity and higher score = more disease activity. Here, Baseline refers to the Baseline of initial studies (EFC11072, ACT11575, EFC10832, SFY13370 and EFC13752).
Time Frame: as for outcome 11
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Sarilumab + Disease Modifying Anti-Rheumatic Drugs (DMARD) | Sarilumab Monotherapy
Number analyzed (Participants) | 1904 | 111
millimeters
  Week 0 | -30.51 (26.78) | -32.30 (27.55)
  Week 4: number analyzed (Participants) | 1887 | 109
  Week 4 | -32.87 (25.60) | -33.63 (25.86)
  Week 8: number analyzed (Participants) | 1863 | 106
  Week 8 | -34.65 (26.25) | -34.25 (25.90)
  Week 12: number analyzed (Participants) | 1830 | 109
  Week 12 | -35.60 (26.77) | -34.24 (28.38)
  Week 24: number analyzed (Participants) | 1785 | 109
  Week 24 | -36.91 (26.50) | -36.12 (27.82)
  Week 36: number analyzed (Participants) | 1729 | 109
  Week 36 | -37.08 (27.18) | -37.13 (24.73)
  Week 48: number analyzed (Participants) | 1674 | 107
  Week 48 | -37.28 (26.93) | -35.98 (28.18)
  Week 60: number analyzed (Participants) | 1622 | 103
  Week 60 | -37.79 (27.38) | -37.82 (25.40)
  Week 72: number analyzed (Participants) | 1589 | 101
  Week 72 | -37.90 (27.26) | -37.95 (26.53)
  Week 84: number analyzed (Participants) | 1552 | 95
  Week 84 | -37.45 (27.82) | -40.52 (26.69)
  Week 96: number analyzed (Participants) | 1512 | 92
  Week 96 | -38.34 (27.34) | -41.46 (26.57)
  Week 120: number analyzed (Participants) | 1459 | 89
  Week 120 | -38.41 (27.43) | -41.67 (26.43)
  Week 144: number analyzed (Participants) | 1394 | 84
  Week 144 | -38.91 (27.52) | -38.52 (26.40)
  Week 168: number analyzed (Participants) | 1328 | 81
  Week 168 | -38.22 (28.26) | -37.27 (27.46)
  Week 192: number analyzed (Participants) | 1267 | 76
  Week 192 | -39.26 (28.16) | -37.79 (32.12)
  Week 216: number analyzed (Participants) | 1191 | 74
  Week 216 | -39.96 (27.72) | -38.72 (32.76)
  Week 240: number analyzed (Participants) | 1133 | 74
  Week 240 | -39.54 (27.79) | -41.64 (30.13)
  Week 264: number analyzed (Participants) | 1061 | 62
  Week 264 | -39.87 (27.31) | -37.84 (32.94)
  Week 288: number analyzed (Participants) | 727 | 26
  Week 288 | -43.68 (25.55) | -48.00 (33.87)
  Week 312: number analyzed (Participants) | 671 | 7
  Week 312 | -44.05 (26.40) | -65.71 (21.40)
  Week 336: number analyzed (Participants) | 543 | 0
  Week 336 | -43.42 (26.95) |
  Week 360: number analyzed (Participants) | 445 | 0
  Week 360 | -44.56 (26.59) |
  Week 384: number analyzed (Participants) | 349 | 0
  Week 384 | -47.19 (26.25) |
  Week 408: number analyzed (Participants) | 214 | 0
  Week 408 | -44.97 (29.16) |
  Week 432: number analyzed (Participants) | 109 | 0
  Week 432 | -49.77 (25.95) |
  Week 456: number analyzed (Participants) | 58 | 0
  Week 456 | -50.40 (24.27) |
  Week 480: number analyzed (Participants) | 43 | 0
  Week 480 | -46.65 (29.66) |
  Week 504: number analyzed (Participants) | 27 | 0
  Week 504 | -48.89 (28.83) |
  Week 516: number analyzed (Participants) | 2 | 0
  Week 516 | -40.50 (36.06) |

23. Secondary Outcome: Change From Baseline in Participant's Assessment of Pain Visual Analogue Scale Score at Week 0, 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240, and 264 of LTS11210
Description: Participants were requested to indicate their pain intensity due to their RA on a 100 mm horizontal VAS, ranging from 0 (no pain) to 100 (worst pain), where a higher score represented more pain due to RA. Here, Baseline refers to the Baseline of initial studies (EFC11072, ACT11575, EFC10832, SFY13370 and EFC13752).
Time Frame: Baseline, Week 0 (post-dose), 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240, and 264 of LTS11210
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Sarilumab + Disease Modifying Anti-Rheumatic Drugs (DMARD) | Sarilumab Monotherapy
Number analyzed (Participants) | 1897 | 111
millimeters
  Week 0 | -31.08 (27.45) | -37.01 (28.73)
  Week 4: number analyzed (Participants) | 1885 | 109
  Week 4 | -34.04 (26.52) | -37.53 (27.28)
  Week 8: number analyzed (Participants) | 1859 | 106
  Week 8 | -35.79 (26.88) | -38.14 (27.16)
  Week 12: number analyzed (Participants) | 1827 | 109
  Week 12 | -36.46 (27.46) | -39.08 (26.79)
  Week 24: number analyzed (Participants) | 1784 | 109
  Week 24 | -37.87 (27.07) | -38.75 (28.12)
  Week 36: number analyzed (Participants) | 1725 | 109
  Week 36 | -37.60 (27.97) | -39.56 (25.72)
  Week 48: number analyzed (Participants) | 1671 | 107
  Week 48 | -38.07 (28.33) | -39.41 (30.12)
  Week 60: number analyzed (Participants) | 1621 | 103
  Week 60 | -38.46 (28.18) | -40.79 (26.20)
  Week 72: number analyzed (Participants) | 1587 | 101
  Week 72 | -38.00 (28.54) | -42.62 (27.33)
  Week 84: number analyzed (Participants) | 1547 | 95
  Week 84 | -38.37 (28.79) | -42.38 (28.69)
  Week 96: number analyzed (Participants) | 1510 | 92
  Week 96 | -38.62 (28.57) | -43.73 (27.59)
  Week 120: number analyzed (Participants) | 1457 | 89
  Week 120 | -39.29 (28.44) | -44.11 (25.69)
  Week 144: number analyzed (Participants) | 1392 | 84
  Week 144 | -39.19 (28.21) | -41.42 (27.31)
  Week 168: number analyzed (Participants) | 1325 | 81
  Week 168 | -39.47 (28.84) | -38.86 (29.46)
  Week 192: number analyzed (Participants) | 1266 | 76
  Week 192 | -40.17 (28.98) | -41.25 (30.44)
  Week 216: number analyzed (Participants) | 1185 | 70
  Week 216 | -40.25 (28.56) | -44.01 (30.27)
  Week 240: number analyzed (Participants) | 1129 | 74
  Week 240 | -40.28 (28.44) | -43.59 (29.22)
  Week 264: number analyzed (Participants) | 1044 | 62
  Week 264 | -41.02 (28.09) | -40.71 (29.79)

24. Secondary Outcome: Change From Baseline in Short Form 36 (SF-36; Version 2) Physical Component Summary (PCS) Score at Week 0, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240 and 264 of LTS11210 - Participants From EFC11072, ACT11575 and EFC10832 Only
Description: SF-36 is a generic 36-item questionnaire consisting of 8 domains, measuring quality of life (QoL) covering 2 summary measures: PCS and mental component summary (MCS). PCS with 4 domains: physical functioning, role limitations due to physical problems, bodily pain, and general health; and MCS with 4 domains: vitality, social functioning, role limitations due to emotional problems, and mental health. Each domain is scored by summing the individual items, which are transformed into a score range from 0 to 100; where 0= worst QoL to 100=best QoL. PCS total score ranged from 0 to 100 with higher scores indicating better physical health. Here, Baseline refers to the Baseline of initial studies (EFC11072, ACT11575, and EFC10832).
Time Frame: Baseline, Week 0 (post-dose), 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240 and 264 of LTS11210
Population: Analysis was performed on safety population. Here, 'overall number of participants analyzed' = participants from studies EFC11072, ACT11575 and EFC10832 evaluable for this outcome measure and 'number analyzed' = participants with available data for each specified category. Data for this outcome measure was not planned to be collected and analyzed for Sarilumab Monotherapy arm, as pre-specified in protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Sarilumab + DMARD: EFC11072, ACT11575 and EFC10832: Participants who completed any of the initial studies: Part A or Part B of EFC11072, ACT11575, and EFC10832 were enrolled in LTS11210 and received sarilumab 150 mg SC qw. Dose could be reduced to 150 mg q2w due to neutropenia, thrombocytopenia or increase in liver enzymes (ALT). After dose regimens selection for Phase 3 studies (150 mg q2w and 200 mg q2w), participants already receiving 150 mg qw were switched to sarilumab 200 mg q2w. Treatment duration per participant was at least 264 weeks from first study drug administration in LTS11210. Participants continued to be treated beyond 264 weeks until sarilumab was commercially available in their respective countries or until 2020, at the latest (maximum duration: 523 weeks). Participants who were already taking concomitant non-biologic DMARDs in initial study continued stable dose of one or combination of conventional synthetic DMARDs they were taking.
Arm/Group | Sarilumab + DMARD: EFC11072, ACT11575 and EFC10832
Number analyzed (Participants) | 1367
units on a scale
  Week 0: number analyzed (Participants) | 1301
  Week 0 | 7.95 (8.29)
  Week 12 | 8.84 (8.45)
  Week 24: number analyzed (Participants) | 1339
  Week 24 | 9.25 (8.59)
  Week 36: number analyzed (Participants) | 1303
  Week 36 | 9.72 (8.85)
  Week 48: number analyzed (Participants) | 1269
  Week 48 | 9.43 (8.89)
  Week 60: number analyzed (Participants) | 1231
  Week 60 | 9.64 (8.53)
  Week 72: number analyzed (Participants) | 1213
  Week 72 | 9.62 (8.78)
  Week 84: number analyzed (Participants) | 1179
  Week 84 | 9.95 (8.97)
  Week 96: number analyzed (Participants) | 1143
  Week 96 | 9.90 (8.90)
  Week 120: number analyzed (Participants) | 1111
  Week 120 | 10.18 (9.12)
  Week 144: number analyzed (Participants) | 1065
  Week 144 | 10.15 (9.18)
  Week 168: number analyzed (Participants) | 1018
  Week 168 | 10.24 (9.24)
  Week 192: number analyzed (Participants) | 967
  Week 192 | 10.34 (9.52)
  Week 216: number analyzed (Participants) | 908
  Week 216 | 10.15 (9.45)
  Week 240: number analyzed (Participants) | 848
  Week 240 | 10.38 (9.21)
  Week 264: number analyzed (Participants) | 754
  Week 264 | 10.32 (9.38)

25. Secondary Outcome: Change From Baseline in Short Form 36 (SF-36; Version 2) Mental Component Summary Score at Week 0, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240 and 264 of LTS11210 - Participants From EFC11072, ACT11575 and EFC10832 Only
Description: SF-36 is a generic 36-item questionnaire consisting of 8 domains, measuring quality of life (QoL) covering 2 summary measures: PCS and MCS. PCS with 4 domains: physical functioning, role limitations due to physical problems, bodily pain, and general health; and MCS with 4 domains: vitality, social functioning, role limitations due to emotional problems, and mental health. Each domain is scored by summing the individual items, which are transformed into a score range from 0 to 100; 0= worst QoL to 100=best QoL. MCS total score ranged from 0 to 100 with higher scores indicating better physical and mental health. Here, Baseline refers to the Baseline of initial studies (EFC11072, ACT11575, and EFC10832).
Time Frame: Baseline, Week 0 (post-dose), 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240 and 264 of LTS11210
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sarilumab + DMARD: EFC11072, ACT11575 and EFC10832
Number analyzed (Participants) | 1367
units on a scale
  Week 0: number analyzed (Participants) | 1301
  Week 0 | 6.43 (10.80)
  Week 12 | 7.15 (11.03)
  Week 24: number analyzed (Participants) | 1339
  Week 24 | 7.43 (11.15)
  Week 36: number analyzed (Participants) | 1303
  Week 36 | 7.20 (11.31)
  Week 48: number analyzed (Participants) | 1269
  Week 48 | 7.48 (11.15)
  Week 60: number analyzed (Participants) | 1231
  Week 60 | 7.43 (11.21)
  Week 72: number analyzed (Participants) | 1213
  Week 72 | 7.25 (11.24)
  Week 84: number analyzed (Participants) | 1179
  Week 84 | 7.29 (11.20)
  Week 96: number analyzed (Participants) | 1143
  Week 96 | 7.47 (11.52)
  Week 120: number analyzed (Participants) | 1111
  Week 120 | 7.69 (11.62)
  Week 144: number analyzed (Participants) | 1065
  Week 144 | 7.22 (11.60)
  Week 168: number analyzed (Participants) | 1018
  Week 168 | 7.29 (11.52)
  Week 192: number analyzed (Participants) | 967
  Week 192 | 7.10 (11.51)
  Week 216: number analyzed (Participants) | 908
  Week 216 | 7.20 (11.91)
  Week 240: number analyzed (Participants) | 848
  Week 240 | 7.23 (12.03)
  Week 264: number analyzed (Participants) | 754
  Week 264 | 7.32 (12.08)

26. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy Fatigue (FACIT-fatigue) Total Score at Week 0, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240 and 264 of LTS11210-Participants From EFC11072, ACT11575 and EFC10832 Only
Description: The FACIT-F is a 13-item questionnaire assessing fatigue where participants scored each item on a 5-point scale (0 to 4): 0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much. The sum of all responses resulted in the FACIT-Fatigue total score ranged from 0 to 52, where higher score = lower level of fatigue and indicates better QoL. A positive change from baseline score indicates an improvement. Here, Baseline refers to the Baseline of initial studies (EFC11072, ACT11575, and EFC10832).
Time Frame: Baseline, Week 0 (post-dose), 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240 and 264 of LTS11210
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sarilumab + DMARD: EFC11072, ACT11575 and EFC10832
Number analyzed (Participants) | 1651
units on a scale
  Week 0: number analyzed (Participants) | 1342
  Week 0 | 9.20 (10.05)
  Week 12 | 10.26 (10.10)
  Week 24: number analyzed (Participants) | 1621
  Week 24 | 10.94 (10.31)
  Week 36: number analyzed (Participants) | 1570
  Week 36 | 10.91 (10.67)
  Week 48: number analyzed (Participants) | 1520
  Week 48 | 10.86 (10.64)
  Week 60: number analyzed (Participants) | 1474
  Week 60 | 10.97 (10.50)
  Week 72: number analyzed (Participants) | 1444
  Week 72 | 10.84 (10.68)
  Week 84: number analyzed (Participants) | 1411
  Week 84 | 10.75 (10.88)
  Week 96: number analyzed (Participants) | 1372
  Week 96 | 11.09 (10.85)
  Week 120: number analyzed (Participants) | 1323
  Week 120 | 11.18 (10.74)
  Week 144: number analyzed (Participants) | 1262
  Week 144 | 11.14 (10.86)
  Week 168: number analyzed (Participants) | 1197
  Week 168 | 11.00 (11.27)
  Week 192: number analyzed (Participants) | 1141
  Week 192 | 10.80 (11.10)
  Week 216: number analyzed (Participants) | 1062
  Week 216 | 11.12 (11.25)
  Week 240: number analyzed (Participants) | 1013
  Week 240 | 11.15 (11.21)
  Week 264: number analyzed (Participants) | 910
  Week 264 | 10.99 (11.19)

27. Secondary Outcome: Change From Baseline in Sleep Visual Analogue Scale Score at Week 0, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240 and 264 of LTS11210 - Participants From EFC11072, and ACT11575 Only
Description: Rheumatoid arthritis (RA), like other chronic illness, is associated with sleep disturbances and is linked to pain, mood, and disease activity. The effect of sarilumab on sleep was assessed on a on 100 mm horizontal VAS scale, ranging from 0 (sleep is not a problem) to 100 (sleep is a major problem), where higher score = more sleep disturbances. Here, Baseline refers to the Baseline of initial studies (EFC11072, and ACT11575).
Time Frame: Baseline, Week 0 (post-dose), 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240 and 264 of LTS11210
Population: Analysis was performed on safety population. Here, 'overall number of participants analyzed' = participants from studies EFC11072, and ACT11575 evaluable for this outcome measure and 'number analyzed' = participants with available data for each specified category. Data for this outcome measure was not planned to be collected and analyzed for Sarilumab Monotherapy arm, as pre-specified in protocol.
Measure: Mean (Standard Deviation); unit: millimeters
Groups:
- Sarilumab + DMARD: EFC11072, and ACT11575: Participants who completed any of the initial studies: Part A or Part B of EFC11072, and ACT11575 were enrolled in LTS11210 and received sarilumab 150 mg SC qw. Dose could be reduced to 150 mg q2w due to neutropenia, thrombocytopenia or increase in liver enzymes (ALT). After dose regimens selection for Phase 3 studies (150 mg q2w and 200 mg q2w), participants already receiving 150 mg qw were switched to sarilumab 200 mg q2w. Treatment duration per participant was at least 264 weeks from first study drug administration in LTS11210. Participants continued to be treated beyond 264 weeks until sarilumab was commercially available in their respective countries or until 2020, at the latest (maximum duration: 523 weeks). Participants who were already taking concomitant non-biologic DMARDs in initial study continued stable dose of one or combination of conventional synthetic DMARDs they were taking.
Arm/Group | Sarilumab + DMARD: EFC11072, and ACT11575
Number analyzed (Participants) | 1231
millimeters
  Week 0: number analyzed (Participants) | 894
  Week 0 | -24.58 (30.96)
  Week 12 | -26.11 (30.59)
  Week 24: number analyzed (Participants) | 1206
  Week 24 | -26.44 (30.94)
  Week 36: number analyzed (Participants) | 1164
  Week 36 | -27.37 (31.52)
  Week 48: number analyzed (Participants) | 1132
  Week 48 | -26.15 (31.37)
  Week 60: number analyzed (Participants) | 1098
  Week 60 | -26.98 (31.24)
  Week 72: number analyzed (Participants) | 1075
  Week 72 | -26.85 (32.16)
  Week 84: number analyzed (Participants) | 1051
  Week 84 | -25.81 (31.90)
  Week 96: number analyzed (Participants) | 1024
  Week 96 | -26.91 (31.63)
  Week 120: number analyzed (Participants) | 983
  Week 120 | -27.63 (32.26)
  Week 144: number analyzed (Participants) | 940
  Week 144 | -26.90 (31.54)
  Week 168: number analyzed (Participants) | 892
  Week 168 | -27.33 (33.25)
  Week 192: number analyzed (Participants) | 853
  Week 192 | -26.87 (32.03)
  Week 216: number analyzed (Participants) | 802
  Week 216 | -28.58 (31.46)
  Week 240: number analyzed (Participants) | 755
  Week 240 | -27.72 (33.07)
  Week 264: number analyzed (Participants) | 705
  Week 264 | -27.71 (32.08)

28. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI): Percent Work Time Missed Due to RA at Week 0, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240 and 264 of LTS11210 - Participants From EFC11072 and ACT11575 Only
Description: WPAI assesses work productivity and impairment. It is 6-item questionnaire used to assess degree to which RA affected work productivity and regular activities over past 7 days. Questions were: Q1 = currently employed; Q2 = hours missed due to RA; Q3 = hours missed due to other reasons; Q4 = hours actually worked; Q5 = degree problem affected productivity while working (0 to 10 scale, with higher numbers indicated less productivity); Q6 = degree problem affected regular activities (0 to 10 scale, with higher numbers indicated greater impairment). The percent work time missed due to RA was a subscale and calculated as: 100*Q2/(Q2+Q4) for those who were currently employed. Subscale score was expressed as impairment percentage (range:0 to 100%) where higher numbers indicate greater impairment and less productivity. Here, Baseline refers to Baseline of initial studies (EFC11072 and ACT11575).
Time Frame: Baseline, Week 0 (post-dose), 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240 and 264 of LTS11210
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sarilumab + DMARD: EFC11072, and ACT11575
Number analyzed (Participants) | 267
units on a scale
  Week 0: number analyzed (Participants) | 191
  Week 0 | -10.82 (30.64)
  Week 12 | -8.62 (28.67)
  Week 24: number analyzed (Participants) | 255
  Week 24 | -11.92 (29.33)
  Week 36: number analyzed (Participants) | 251
  Week 36 | -9.62 (30.08)
  Week 48: number analyzed (Participants) | 243
  Week 48 | -11.39 (29.92)
  Week 60: number analyzed (Participants) | 236
  Week 60 | -10.03 (25.74)
  Week 72: number analyzed (Participants) | 216
  Week 72 | -9.10 (28.14)
  Week 84: number analyzed (Participants) | 206
  Week 84 | -8.20 (27.06)
  Week 96: number analyzed (Participants) | 209
  Week 96 | -11.32 (30.28)
  Week 120: number analyzed (Participants) | 189
  Week 120 | -8.62 (32.95)
  Week 144: number analyzed (Participants) | 183
  Week 144 | -9.01 (30.16)
  Week 168: number analyzed (Participants) | 176
  Week 168 | -10.38 (31.48)
  Week 192: number analyzed (Participants) | 166
  Week 192 | -8.99 (29.24)
  Week 216: number analyzed (Participants) | 147
  Week 216 | -11.17 (29.35)
  Week 240: number analyzed (Participants) | 147
  Week 240 | -8.57 (26.11)
  Week 264: number analyzed (Participants) | 133
  Week 264 | -13.40 (30.57)

29. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment: Percent Impairment While Working Due to RA at Weeks 0, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240 and 264 of LTS11210 - Participants From EFC11072, and ACT11575 Only
Description: WPAI assesses work productivity and impairment. It is 6-item questionnaire used to assess degree to which RA affected work productivity and regular activities over past 7 days. Questions were: Q1 = currently employed; Q2 = hours missed due to RA; Q3 = hours missed due to other reasons; Q4 = hours actually worked; Q5 = degree problem affected productivity while working (0 to 10 scale, with higher numbers = less productivity); Q6 = degree problem affected regular activities (0 to 10 scale, with higher numbers = greater impairment). Percentage impairment while working due to RA was subscale and calculated as: 10*Q5 for those who were currently employed and actually worked in past 7 days. Subscale score=expressed as impairment percentage (range:0 to 100%), where higher numbers=greater impairment and less productivity. Here, Baseline refers to the Baseline of initial studies (EFC11072 and ACT11575).
Time Frame: Baseline, Weeks 0 (post-dose), 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240 and 264 of LTS11210
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sarilumab + DMARD: EFC11072, and ACT11575
Number analyzed (Participants) | 273
units on a scale
  Week 0: number analyzed (Participants) | 194
  Week 0 | -21.65 (27.74)
  Week 12 | -22.16 (26.53)
  Week 24: number analyzed (Participants) | 258
  Week 24 | -23.45 (26.70)
  Week 36: number analyzed (Participants) | 254
  Week 36 | -27.01 (27.11)
  Week 48: number analyzed (Participants) | 252
  Week 48 | -24.76 (26.05)
  Week 60: number analyzed (Participants) | 240
  Week 60 | -25.17 (25.12)
  Week 72: number analyzed (Participants) | 224
  Week 72 | -24.33 (27.57)
  Week 84: number analyzed (Participants) | 214
  Week 84 | -24.02 (27.09)
  Week 96: number analyzed (Participants) | 212
  Week 96 | -26.42 (27.11)
  Week 120: number analyzed (Participants) | 189
  Week 120 | -24.02 (27.63)
  Week 144: number analyzed (Participants) | 184
  Week 144 | -24.67 (28.20)
  Week 168: number analyzed (Participants) | 181
  Week 168 | -24.25 (28.46)
  Week 192: number analyzed (Participants) | 168
  Week 192 | -25.24 (26.60)
  Week 216: number analyzed (Participants) | 147
  Week 216 | -24.56 (27.28)
  Week 240: number analyzed (Participants) | 155
  Week 240 | -24.39 (26.48)
  Week 264: number analyzed (Participants) | 135
  Week 264 | -25.26 (27.40)

30. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment: Percent Overall Work Impairment Due to RA at Weeks 0, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240 and 264 of LTS11210 - Participants From EFC11072, and ACT11575 Only
Description: WPAI assesses work productivity and impairment. It is 6-item questionnaire used to assess degree to which RA affected work productivity and regular activities over past 7 days. Questions were: Q1 = currently employed; Q2 = hours missed due to RA; Q3 = hours missed due to other reasons; Q4 = hours actually worked; Q5 = degree problem affected productivity while working (0 to 10 scale, with higher numbers indicated less productivity); Q6 = degree problem affected regular activities (0 10 scale, with higher numbers indicated greater impairment). Percent overall work impairment due to RA was subscale and calculated as: 100*Q2/(Q2+Q4)+100*[(1- Q2/(Q2+Q4))*(Q5/10)] for those who were currently employed . Subscale score = expressed as impairment percentage (range: 0 to 100%) where higher numbers indicate greater impairment. Here, Baseline refers to Baseline of initial studies (EFC11072 and ACT11575).
Time Frame: Baseline, Weeks 0 (post-dose), 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240 and 264 of LTS11210
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sarilumab + DMARD: EFC11072, and ACT11575
Number analyzed (Participants) | 246
units on a scale
  Week 0: number analyzed (Participants) | 172
  Week 0 | -22.84 (30.73)
  Week 12 | -23.13 (27.98)
  Week 24: number analyzed (Participants) | 232
  Week 24 | -25.39 (28.84)
  Week 36: number analyzed (Participants) | 230
  Week 36 | -28.13 (29.01)
  Week 48: number analyzed (Participants) | 223
  Week 48 | -24.72 (29.38)
  Week 60: number analyzed (Participants) | 222
  Week 60 | -26.44 (28.03)
  Week 72: number analyzed (Participants) | 200
  Week 72 | -25.06 (29.84)
  Week 84: number analyzed (Participants) | 193
  Week 84 | -23.62 (29.25)
  Week 96: number analyzed (Participants) | 193
  Week 96 | -27.06 (30.60)
  Week 120: number analyzed (Participants) | 172
  Week 120 | -24.15 (31.14)
  Week 144: number analyzed (Participants) | 168
  Week 144 | -23.97 (32.05)
  Week 168: number analyzed (Participants) | 162
  Week 168 | -24.59 (31.16)
  Week 192: number analyzed (Participants) | 155
  Week 192 | -24.77 (29.63)
  Week 216: number analyzed (Participants) | 136
  Week 216 | -24.54 (31.55)
  Week 240: number analyzed (Participants) | 140
  Week 240 | -25.05 (29.26)
  Week 264: number analyzed (Participants) | 122
  Week 264 | -27.10 (28.75)

31. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment: Percent Activity Impairment Due to RA at Weeks 0, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240 and 264 of LTS11210 - Participants From EFC11072, and ACT11575 Only
Description: WPAI assesses work productivity and impairment. It is 6-item questionnaire used to assess degree to which RA affected work productivity and regular activities over past 7 days. Questions were: Q1 = currently employed; Q2 = hours missed due to RA; Q3 = hours missed due to other reasons; Q4 = hours actually worked; Q5 = degree problem affected productivity while working (0 to 10 scale, with higher numbers indicated less productivity); Q6 = degree problem affected regular activities (0 10 scale, with higher numbers indicated greater impairment). Percent activity impairment due to RA was a subscale and calculated as: 10*Q6 for all respondents. Subscale score=expressed as impairment percentage (range: 0 to 100%) where higher numbers indicate greater impairment. Here, Baseline refers to Baseline of initial studies (EFC11072 and ACT11575).
Time Frame: Baseline, Weeks 0 (post-dose), 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240 and 264 of LTS11210
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sarilumab + DMARD: EFC11072, and ACT11575
Number analyzed (Participants) | 1157
units on a scale
  Week 0: number analyzed (Participants) | 846
  Week 0 | -26.47 (29.30)
  Week 12 | -28.02 (27.44)
  Week 24: number analyzed (Participants) | 1121
  Week 24 | -28.76 (27.62)
  Week 36: number analyzed (Participants) | 1095
  Week 36 | -29.71 (28.03)
  Week 48: number analyzed (Participants) | 1061
  Week 48 | -29.11 (28.28)
  Week 60: number analyzed (Participants) | 1034
  Week 60 | -29.81 (27.78)
  Week 72: number analyzed (Participants) | 1013
  Week 72 | -29.61 (29.02)
  Week 84: number analyzed (Participants) | 985
  Week 84 | -30.28 (29.53)
  Week 96: number analyzed (Participants) | 954
  Week 96 | -30.28 (28.32)
  Week 120: number analyzed (Participants) | 924
  Week 120 | -30.42 (28.78)
  Week 144: number analyzed (Participants) | 883
  Week 144 | -30.29 (28.90)
  Week 168: number analyzed (Participants) | 840
  Week 168 | -30.64 (29.30)
  Week 192: number analyzed (Participants) | 804
  Week 192 | -30.88 (29.36)
  Week 216: number analyzed (Participants) | 753
  Week 216 | -30.36 (29.34)
  Week 240: number analyzed (Participants) | 722
  Week 240 | -31.12 (29.63)
  Week 264: number analyzed (Participants) | 645
  Week 264 | -31.97 (28.77)

32. Secondary Outcome: Change From Baseline in Work Productivity Survey - Rheumatoid Arthritis (WPS-RA) at Weeks 0, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240 and 264 of LTS11210: Work Days Missed Due to Arthritis - Participants From EFC10832 Only
Description: The WPS-RA is a validated questionnaire that evaluates productivity limitations within work and within home associated with arthritis over the previous month. The questionnaire was interviewer-administered and was based on participant self-report. It contains 9 questions addressing employment status (1 item), productivity at work (3 items), and within and outside the home (5 items). Change from Baseline in number of work days missed in the last month due to arthritis by the participant was reported in the outcome measure. Here, Baseline refers to the Baseline of initial study (EFC10832).
Time Frame: Baseline, Weeks 0 (post-dose), 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240 and 264 of LTS11210
Population: Analysis was performed on safety population. Here, 'overall number of participants analyzed' = participants from study EFC10832 evaluable for this outcome measure and 'number analyzed' = participants with available data for each specified category. Data for this outcome measure was not planned to be collected and analyzed for Sarilumab Monotherapy arm, as pre-specified in protocol.
Measure: Mean (Standard Deviation); unit: days
Groups:
- Sarilumab + DMARD: EFC10832: Participants who completed study EFC10832 were enrolled in LTS11210 and received sarilumab 150 mg SC qw. Dose could be reduced to 150 mg q2w due to neutropenia, thrombocytopenia or increase in liver enzymes (ALT). After dose regimens selection for Phase 3 studies (150 mg q2w and 200 mg q2w), participants already receiving 150 mg qw were switched to sarilumab 200 mg q2w. Treatment duration per participant was at least 264 weeks from first study drug administration in LTS11210. Participants continued to be treated beyond 264 weeks until sarilumab was commercially available in their respective countries or until 2020, at the latest (maximum duration: 523 weeks). Participants who were already taking concomitant non-biologic DMARDs in initial study continued stable dose of one or combination of conventional synthetic DMARDs they were taking.
Arm/Group | Sarilumab + DMARD: EFC10832
Number analyzed (Participants) | 145
days
  Week 0 | -2.72 (6.38)
  Week 12: number analyzed (Participants) | 127
  Week 12 | -3.66 (6.80)
  Week 24: number analyzed (Participants) | 125
  Week 24 | -3.70 (6.85)
  Week 36: number analyzed (Participants) | 121
  Week 36 | -3.73 (7.08)
  Week 48: number analyzed (Participants) | 116
  Week 48 | -3.37 (7.18)
  Week 60: number analyzed (Participants) | 114
  Week 60 | -3.55 (6.93)
  Week 72: number analyzed (Participants) | 111
  Week 72 | -3.58 (7.07)
  Week 84: number analyzed (Participants) | 106
  Week 84 | -3.11 (8.49)
  Week 96: number analyzed (Participants) | 101
  Week 96 | -3.47 (7.57)
  Week 120: number analyzed (Participants) | 101
  Week 120 | -3.54 (7.56)
  Week 144: number analyzed (Participants) | 94
  Week 144 | -3.51 (6.84)
  Week 168: number analyzed (Participants) | 88
  Week 168 | -3.73 (7.37)
  Week 192: number analyzed (Participants) | 80
  Week 192 | -3.76 (7.21)
  Week 216: number analyzed (Participants) | 74
  Week 216 | -3.51 (7.30)
  Week 240: number analyzed (Participants) | 73
  Week 240 | -2.44 (6.70)
  Week 264: number analyzed (Participants) | 66
  Week 264 | -2.86 (5.83)

33. Secondary Outcome: Change From Baseline in WPS-RA at Weeks 0, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240 and 264 of LTS11210: Days With Work Productivity Reduced by >=50% Due to Arthritis - Participants From EFC10832 Only
Description: The WPS-RA is a validated questionnaire that evaluates productivity limitations within work and within home associated with RA over the previous month. The questionnaire was interviewer-administered and was based on participant self-report. It contains 9 questions addressing employment status (1 item), productivity at work (3 items), and within and outside the home (5 items). Change from Baseline in number of work days with reduced productivity by >= 50% in the last month by the participant was reported in the outcome measure. Here, Baseline refers to the Baseline of initial study (EFC10832).
Time Frame: Baseline, Weeks 0 (post-dose), 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240 and 264 of LTS11210
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Sarilumab + DMARD: EFC10832
Number analyzed (Participants) | 145
days
  Week 0 | -3.47 (7.64)
  Week 12: number analyzed (Participants) | 126
  Week 12 | -4.93 (9.22)
  Week 24: number analyzed (Participants) | 123
  Week 24 | -5.14 (7.67)
  Week 36: number analyzed (Participants) | 122
  Week 36 | -5.47 (8.41)
  Week 48: number analyzed (Participants) | 115
  Week 48 | -5.75 (8.14)
  Week 60: number analyzed (Participants) | 114
  Week 60 | -5.16 (7.96)
  Week 72: number analyzed (Participants) | 110
  Week 72 | -5.21 (7.74)
  Week 84: number analyzed (Participants) | 105
  Week 84 | -4.40 (8.27)
  Week 96: number analyzed (Participants) | 101
  Week 96 | -5.03 (6.91)
  Week 120: number analyzed (Participants) | 101
  Week 120 | -4.63 (7.47)
  Week 144: number analyzed (Participants) | 94
  Week 144 | -4.88 (7.53)
  Week 168: number analyzed (Participants) | 88
  Week 168 | -4.67 (7.06)
  Week 192: number analyzed (Participants) | 80
  Week 192 | -4.55 (7.25)
  Week 216: number analyzed (Participants) | 74
  Week 216 | -4.42 (8.01)
  Week 240: number analyzed (Participants) | 73
  Week 240 | -3.48 (7.56)
  Week 264: number analyzed (Participants) | 66
  Week 264 | -3.97 (5.02)

34. Secondary Outcome: Change From Baseline in WPS-RA at Weeks 0, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240 and 264 of LTS11210: Arthritis Interference With Work Productivity - Participants From EFC10832 Only
Description: The WPS-RA is a validated questionnaire that evaluates productivity limitations within work and within home associated with RA over the previous month. The questionnaire was interviewer-administered and was based on participant self-report. It contains 9 questions addressing employment status (1 item), productivity at work (3 items), and within and outside the home (5 items). Interference in the last month with work productivity was measured on a scale that ranged from 0 (no interference) to 10 (complete interference), where higher scores indicated more interference. Here, Baseline refers to the Baseline of initial study (EFC10832).
Time Frame: Baseline, Weeks 0 (post-dose), 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240 and 264 of LTS11210
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sarilumab + DMARD: EFC10832
Number analyzed (Participants) | 144
units on a scale
  Week 0 | -20.83 (30.51)
  Week 12: number analyzed (Participants) | 127
  Week 12 | -27.95 (58.67)
  Week 24: number analyzed (Participants) | 124
  Week 24 | -35.16 (31.45)
  Week 36: number analyzed (Participants) | 123
  Week 36 | -37.48 (33.72)
  Week 48: number analyzed (Participants) | 115
  Week 48 | -36.78 (31.58)
  Week 60: number analyzed (Participants) | 115
  Week 60 | -40.35 (33.19)
  Week 72: number analyzed (Participants) | 111
  Week 72 | -38.74 (32.73)
  Week 84: number analyzed (Participants) | 106
  Week 84 | -39.62 (41.56)
  Week 96: number analyzed (Participants) | 102
  Week 96 | -42.35 (32.19)
  Week 120: number analyzed (Participants) | 102
  Week 120 | -37.84 (32.32)
  Week 144: number analyzed (Participants) | 95
  Week 144 | -39.16 (32.28)
  Week 168: number analyzed (Participants) | 90
  Week 168 | -38.11 (32.25)
  Week 192: number analyzed (Participants) | 81
  Week 192 | -40.74 (34.96)
  Week 216: number analyzed (Participants) | 74
  Week 216 | -39.19 (37.00)
  Week 240: number analyzed (Participants) | 73
  Week 240 | -38.22 (38.24)
  Week 264: number analyzed (Participants) | 66
  Week 264 | -39.24 (36.09)

35. Secondary Outcome: Change From Baseline in WPS-RA at Weeks 0, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240 and 264 of LTS11210: House Work Days Missed Due to Arthritis - Participants From EFC10832 Only
Description: 'The WPS-RA is a validated questionnaire that evaluates productivity limitations within work and within home associated with RA over the previous month. The questionnaire was interviewer-administered and was based on participant self-report. It contains 9 questions addressing employment status (1 item), productivity at work (3 items), and within and outside the home (5 items). Change from baseline in number of days with no household work/household work missed in the last month by the participants was reported. Here, Baseline refers to the Baseline of initial study (EFC10832).
Time Frame: Baseline, Weeks 0 (post-dose), 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240 and 264 of LTS11210
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Sarilumab + DMARD: EFC10832
Number analyzed (Participants) | 446
days
  Week 0 | -4.65 (9.44)
  Week 12: number analyzed (Participants) | 401
  Week 12 | -6.17 (10.29)
  Week 24: number analyzed (Participants) | 397
  Week 24 | -6.55 (9.92)
  Week 36: number analyzed (Participants) | 388
  Week 36 | -6.65 (10.36)
  Week 48: number analyzed (Participants) | 373
  Week 48 | -6.61 (10.57)
  Week 60: number analyzed (Participants) | 364
  Week 60 | -6.84 (10.47)
  Week 72: number analyzed (Participants) | 355
  Week 72 | -6.50 (10.72)
  Week 84: number analyzed (Participants) | 343
  Week 84 | -6.56 (10.63)
  Week 96: number analyzed (Participants) | 336
  Week 96 | -6.80 (10.32)
  Week 120: number analyzed (Participants) | 323
  Week 120 | -6.81 (10.31)
  Week 144: number analyzed (Participants) | 309
  Week 144 | -6.78 (10.67)
  Week 168: number analyzed (Participants) | 283
  Week 168 | -7.04 (10.13)
  Week 192: number analyzed (Participants) | 274
  Week 192 | -6.74 (10.51)
  Week 216: number analyzed (Participants) | 261
  Week 216 | -6.78 (10.07)
  Week 240: number analyzed (Participants) | 243
  Week 240 | -6.82 (10.02)
  Week 264: number analyzed (Participants) | 230
  Week 264 | -6.95 (10.16)

36. Secondary Outcome: Change From Baseline in WPS-RA at Weeks 0, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240 and 264 of LTS11210: Days With Household Work Productivity Reduced by >=50% Due to Arthritis - Participants From EFC10832 Only
Description: The WPS-RA is a validated questionnaire that evaluates productivity limitations within work and within home associated with RA over the previous month. The questionnaire was interviewer-administered and was based on participant self-report. It contains 9 questions addressing employment status (1 item), productivity at work (3 items), and within and outside the home (5 items). Change from baseline in number of days with reduced household work productivity by >= 50% in the last month by the participants was reported. Here, Baseline refers to the Baseline of initial study (EFC10832).
Time Frame: Baseline, Weeks 0 (post-dose), 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240 and 264 of LTS11210
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Sarilumab + DMARD: EFC10832
Number analyzed (Participants) | 445
days
  Week 0 | -4.08 (10.24)
  Week 12: number analyzed (Participants) | 402
  Week 12 | -5.64 (10.93)
  Week 24: number analyzed (Participants) | 395
  Week 24 | -6.01 (10.40)
  Week 36: number analyzed (Participants) | 387
  Week 36 | -6.57 (10.29)
  Week 48: number analyzed (Participants) | 372
  Week 48 | -7.06 (10.13)
  Week 60: number analyzed (Participants) | 363
  Week 60 | -7.01 (10.30)
  Week 72: number analyzed (Participants) | 353
  Week 72 | -6.70 (10.72)
  Week 84: number analyzed (Participants) | 342
  Week 84 | -6.38 (10.79)
  Week 96: number analyzed (Participants) | 334
  Week 96 | -7.05 (10.62)
  Week 120: number analyzed (Participants) | 322
  Week 120 | -7.12 (10.37)
  Week 144: number analyzed (Participants) | 308
  Week 144 | -6.58 (10.59)
  Week 168: number analyzed (Participants) | 284
  Week 168 | -6.39 (10.28)
  Week 192: number analyzed (Participants) | 274
  Week 192 | -6.01 (10.07)
  Week 216: number analyzed (Participants) | 259
  Week 216 | -6.27 (10.30)
  Week 240: number analyzed (Participants) | 241
  Week 240 | -6.31 (9.99)
  Week 264: number analyzed (Participants) | 229
  Week 264 | -6.93 (9.43)

37. Secondary Outcome: Change From Baseline in WPS-RA at Weeks 0, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240 and 264 of LTS11210: Days With Family/Social/Leisure Activities Missed Due to Arthritis - Participants From EFC10832 Only
Description: The WPS-RA is a validated questionnaire that evaluates productivity limitations within work and within home associated with RA over the previous month. The questionnaire was interviewer-administered and was based on participant self-report. It contains 9 questions addressing employment status (1 item), productivity at work (3 items), and within and outside the home (5 items). Change from baseline in number of days missed of family/social/leisure activities in the last month by the participants was reported. Here, Baseline refers to the Baseline of initial study (EFC10832).
Time Frame: Baseline, Weeks 0 (post-dose), 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240 and 264 of LTS11210
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Sarilumab + DMARD: EFC10832
Number analyzed (Participants) | 447
days
  Week 0 | -2.94 (8.34)
  Week 12: number analyzed (Participants) | 401
  Week 12 | -4.16 (8.38)
  Week 24: number analyzed (Participants) | 397
  Week 24 | -4.50 (8.42)
  Week 36: number analyzed (Participants) | 388
  Week 36 | -4.38 (8.88)
  Week 48: number analyzed (Participants) | 373
  Week 48 | -4.44 (8.51)
  Week 60: number analyzed (Participants) | 364
  Week 60 | -4.46 (8.31)
  Week 72: number analyzed (Participants) | 354
  Week 72 | -4.20 (8.52)
  Week 84: number analyzed (Participants) | 343
  Week 84 | -4.31 (8.30)
  Week 96: number analyzed (Participants) | 335
  Week 96 | -4.38 (8.03)
  Week 120: number analyzed (Participants) | 323
  Week 120 | -4.43 (8.01)
  Week 144: number analyzed (Participants) | 309
  Week 144 | -4.17 (7.90)
  Week 168: number analyzed (Participants) | 285
  Week 168 | -4.12 (8.16)
  Week 192: number analyzed (Participants) | 272
  Week 192 | -4.23 (8.17)
  Week 216: number analyzed (Participants) | 261
  Week 216 | -3.93 (8.03)
  Week 240: number analyzed (Participants) | 242
  Week 240 | -4.03 (8.26)
  Week 264: number analyzed (Participants) | 230
  Week 264 | -3.85 (7.65)

38. Secondary Outcome: Change From Baseline in WPS-RA at Weeks 0, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240 and 264 of LTS11210: Days With Outside Help Hired Due to Arthritis- Participants From EFC10832 Only
Description: The WPS-RA is a validated questionnaire that evaluates productivity limitations within work and within home associated with RA over the previous month. The questionnaire was interviewer-administered and was based on participant self-report. It contains 9 questions addressing employment status (1 item), productivity at work (3 items), and within and outside the home (5 items). Change from baseline in number of days with outside help hired in the last month by the participant was reported. Here, Baseline refers to the Baseline of initial study (EFC10832).
Time Frame: Baseline, Weeks 0 (post-dose), 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240 and 264 of LTS11210
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Sarilumab + DMARD: EFC10832
Number analyzed (Participants) | 446
days
  Week 0 | -2.92 (10.14)
  Week 12: number analyzed (Participants) | 401
  Week 12 | -4.24 (10.16)
  Week 24: number analyzed (Participants) | 397
  Week 24 | -4.12 (10.47)
  Week 36: number analyzed (Participants) | 388
  Week 36 | -4.28 (10.27)
  Week 48: number analyzed (Participants) | 373
  Week 48 | -4.58 (10.12)
  Week 60: number analyzed (Participants) | 364
  Week 60 | -4.21 (10.16)
  Week 72: number analyzed (Participants) | 354
  Week 72 | -4.00 (9.52)
  Week 84: number analyzed (Participants) | 343
  Week 84 | -3.81 (9.67)
  Week 96: number analyzed (Participants) | 335
  Week 96 | -3.90 (10.11)
  Week 120: number analyzed (Participants) | 323
  Week 120 | -3.90 (9.62)
  Week 144: number analyzed (Participants) | 309
  Week 144 | -3.91 (9.73)
  Week 168: number analyzed (Participants) | 285
  Week 168 | -4.14 (10.00)
  Week 192: number analyzed (Participants) | 273
  Week 192 | -3.93 (10.14)
  Week 216: number analyzed (Participants) | 261
  Week 216 | -4.19 (9.84)
  Week 240: number analyzed (Participants) | 242
  Week 240 | -4.12 (10.43)
  Week 264: number analyzed (Participants) | 230
  Week 264 | -4.05 (9.67)

39. Secondary Outcome: Change From Baseline in WPS-RA at Weeks 0, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240 and 264 of LTS11210: Arthritis Interference With Household Work Productivity - Participants From EFC10832 Only
Description: The WPS-RA is a validated questionnaire that evaluates productivity limitations within work and within home associated with RA over the previous month. The questionnaire was interviewer-administered and was based on participant self-report. It contains 9 questions addressing employment status (1 item), productivity at work (3 items), and within and outside the home (5 items). The RA interference in the last month with household work productivity was measured on a scale that ranged from 0 (no interference) to 10 (complete interference), where higher scores indicated more interference. Here, Baseline refers to the Baseline of initial study (EFC10832).
Time Frame: Baseline, Weeks 0 (post-dose), 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192, 216, 240 and 264 of LTS11210
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sarilumab + DMARD: EFC10832
Number analyzed (Participants) | 444
units on a scale
  Week 0 | -23.24 (35.09)
  Week 12: number analyzed (Participants) | 401
  Week 12 | -33.49 (35.76)
  Week 24: number analyzed (Participants) | 399
  Week 24 | -36.94 (36.75)
  Week 36: number analyzed (Participants) | 388
  Week 36 | -36.42 (39.35)
  Week 48: number analyzed (Participants) | 373
  Week 48 | -37.45 (34.85)
  Week 60: number analyzed (Participants) | 365
  Week 60 | -38.19 (34.55)
  Week 72: number analyzed (Participants) | 355
  Week 72 | -36.48 (35.37)
  Week 84: number analyzed (Participants) | 344
  Week 84 | -35.61 (39.69)
  Week 96: number analyzed (Participants) | 335
  Week 96 | -36.81 (36.04)
  Week 120: number analyzed (Participants) | 324
  Week 120 | -38.86 (35.22)
  Week 144: number analyzed (Participants) | 310
  Week 144 | -36.23 (37.52)
  Week 168: number analyzed (Participants) | 286
  Week 168 | -36.01 (39.84)
  Week 192: number analyzed (Participants) | 274
  Week 192 | -35.80 (40.99)
  Week 216: number analyzed (Participants) | 260
  Week 216 | -38.54 (39.81)
  Week 240: number analyzed (Participants) | 240
  Week 240 | -40.08 (35.68)
  Week 264: number analyzed (Participants) | 228
  Week 264 | -38.07 (42.39)

40. Secondary Outcome: Sub-study: Number of Participants Who Reported Adverse Events Related to Pre-filled Syringe With Safety System
Description: AEs related to PFS-S included PTC-related AEs, device-related AEs, or AEs of injection site reaction. In this outcome measure, only PTC-related AEs, device-related AEs, or AEs of injection site reaction assessed during the sub-study were reported. TEAEs and SAEs reported during the sub-study were included in the main study data and no separate data collection and analysis was performed, as pre-planned in the protocol .
Time Frame: From Week 24 to 36
Population: Analysis was performed on all participants who were enrolled in the sub-study.
Measure: Count of Participants; unit: Participants
Arm/Group | PFS-S Sarilumab 150 mg q2w | PFS-S Sarilumab 200 mg q2w | PFS-S Sarilumab 200 to 150 mg q2w
Number analyzed (Participants) | 25 | 98 | 1
Participants
  PTC-related AEs | 0 | 0 | 0
  Device-related AEs | 0 | 0 | 0
  AEs of injection site reaction | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose (i.e., Day 1 of study LTS11210) of IMP to last dose of IMP + 60 days (maximum duration: up to 523 weeks)
Description: Reported AEs and deaths were TEAEs that developed/worsened in grade or became serious during TEAE period (defined as the time from the first dose of the IMP to the last dose of IMP + 60 days). As pre-specified and initially planned, TEAEs and SAEs reported during the sub-study were included in the main study data and no separate analysis was done. Analysis was performed on safety population.
Arm/Group | Sarilumab + Disease Modifying Anti-Rheumatic Drugs (DMARD) | Sarilumab Monotherapy
All-Cause Mortality (participants affected / at risk) | 49/1910 | 3/111
Serious Adverse Events (participants affected / at risk) | 617/1910 | 27/111
Other Adverse Events (participants affected / at risk) | 1444/1910 | 82/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sarilumab + Disease Modifying Anti-Rheumatic Drugs (DMARD) (N=1910) | Sarilumab Monotherapy (N=111)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Anaemia Megaloblastic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Blood Loss Anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Bone Marrow Failure (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphatic Insufficiency (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 11 (12) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Spontaneous Haemorrhage (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Acute Coronary Syndrome (Cardiac disorders) | 2 (2) | 0 (0)
Acute Left Ventricular Failure (Cardiac disorders) | 1 (1) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 11 (11) | 0 (0)
Angina Pectoris (Cardiac disorders) | 3 (3) | 0 (0)
Angina Unstable (Cardiac disorders) | 2 (2) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 9 (11) | 2 (3)
Atrial Flutter (Cardiac disorders) | 3 (4) | 0 (0)
Atrial Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular Block Complete (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac Failure (Cardiac disorders) | 4 (4) | 0 (0)
Cardiac Failure Acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac Tamponade (Cardiac disorders) | 2 (2) | 0 (0)
Cardio-Respiratory Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiogenic Shock (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary Failure (Cardiac disorders) | 2 (2) | 0 (0)
Congestive Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 3 (3) | 0 (0)
Coronary Artery Perforation (Cardiac disorders) | 1 (1) | 0 (0)
Coronary Artery Stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Left Ventricular Failure (Cardiac disorders) | 1 (1) | 1 (1)
Microvascular Coronary Artery Disease (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 5 (5) | 0 (0)
Myocardial Ischaemia (Cardiac disorders) | 4 (4) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Sinus Node Dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular Asystole (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 2 (2) | 0 (0)
Thyroiditis (Endocrine disorders) | 1 (1) | 0 (0)
Thyroiditis Subacute (Endocrine disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 4 (4) | 0 (0)
Central Vision Loss (Eye disorders) | 1 (1) | 0 (0)
Choroiditis (Eye disorders) | 1 (1) | 0 (0)
Dry Age-Related Macular Degeneration (Eye disorders) | 1 (1) | 0 (0)
Macular Hole (Eye disorders) | 1 (1) | 0 (0)
Neovascular Age-Related Macular Degeneration (Eye disorders) | 1 (1) | 0 (0)
Optic Ischaemic Neuropathy (Eye disorders) | 1 (1) | 0 (0)
Retinal Vascular Thrombosis (Eye disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Appendicolith (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chronic Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Crohn's Disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diverticular Perforation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diverticulum Intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum Intestinal Haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterovesical Fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Femoral Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric Ulcer Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastrointestinal Inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hernial Eventration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus Hernia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Ileal Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Incarcerated Umbilical Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inflammatory Bowel Disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Intestinal Dilatation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 3 (3) | 0 (0)
Irritable Bowel Syndrome (Gastrointestinal disorders) | 2 (2) | 0 (0)
Large Intestine Perforation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Noninfectious Peritonitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic Necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic Pseudocyst Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatitis Acute (Gastrointestinal disorders) | 5 (5) | 0 (0)
Pancreatitis Necrotising (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritoneal Adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal Haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Rectal Prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 2 (5) | 0 (0)
Umbilical Hernia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cardiac Death (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Multiple Organ Dysfunction Syndrome (General disorders) | 3 (3) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 6 (6) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Sudden Death (General disorders) | 1 (1) | 0 (0)
Bile Duct Stone (Hepatobiliary disorders) | 3 (3) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 9 (9) | 0 (0)
Cholecystitis Acute (Hepatobiliary disorders) | 3 (3) | 1 (1)
Cholecystitis Chronic (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 24 (24) | 0 (0)
Cholelithiasis Obstructive (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portosplenomesenteric Venous Thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abdominal Abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess Limb (Infections and infestations) | 6 (6) | 0 (0)
Abscess Neck (Infections and infestations) | 1 (1) | 0 (0)
Abscess Oral (Infections and infestations) | 1 (1) | 0 (0)
Abscess Soft Tissue (Infections and infestations) | 2 (2) | 0 (0)
Acute Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Anal Abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 4 (4) | 0 (0)
Arteriovenous Graft Site Infection (Infections and infestations) | 1 (1) | 0 (0)
Arthritis Bacterial (Infections and infestations) | 6 (7) | 1 (1)
Arthritis Infective (Infections and infestations) | 1 (1) | 0 (0)
Atypical Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bacterial Dacryocystitis (Infections and infestations) | 1 (1) | 0 (0)
Bartholin's Abscess (Infections and infestations) | 1 (1) | 0 (0)
Bone Tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 4 (4) | 0 (0)
Bronchitis Fungal (Infections and infestations) | 1 (1) | 0 (0)
Bullous Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Bursitis Infective (Infections and infestations) | 2 (2) | 0 (0)
Covid-19 Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Carbuncle (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 21 (24) | 0 (0)
Cellulitis Staphylococcal (Infections and infestations) | 3 (3) | 0 (0)
Cholecystitis Infective (Infections and infestations) | 1 (1) | 0 (0)
Clostridium Difficile Infection (Infections and infestations) | 1 (1) | 2 (2)
Coccidioidomycosis (Infections and infestations) | 1 (1) | 0 (0)
Colonic Abscess (Infections and infestations) | 2 (2) | 0 (0)
Dengue Fever (Infections and infestations) | 1 (1) | 0 (0)
Device Related Infection (Infections and infestations) | 1 (1) | 0 (0)
Diarrhoea Infectious (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 7 (7) | 1 (1)
Endocarditis (Infections and infestations) | 2 (2) | 0 (0)
Endometritis (Infections and infestations) | 1 (1) | 0 (0)
Enteritis Infectious (Infections and infestations) | 1 (1) | 0 (0)
Epiglottitis (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 5 (5) | 0 (0)
Escherichia Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Extradural Abscess (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gas Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis Bacterial (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis Salmonella (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 1 (1) | 0 (0)
Haematoma Infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes Ophthalmic (Infections and infestations) | 1 (1) | 0 (0)
Herpes Zoster (Infections and infestations) | 5 (5) | 1 (1)
Histoplasmosis Disseminated (Infections and infestations) | 1 (1) | 0 (0)
Infected Bite (Infections and infestations) | 1 (1) | 0 (0)
Infected Skin Ulcer (Infections and infestations) | 6 (6) | 0 (0)
Infectious Pleural Effusion (Infections and infestations) | 2 (2) | 0 (0)
Infective Exacerbation Of Bronchiectasis (Infections and infestations) | 2 (2) | 0 (0)
Infective Exacerbation Of Chronic Obstructive Airways Disease (Infections and infestations) | 2 (2) | 0 (0)
Large Intestine Infection (Infections and infestations) | 1 (2) | 0 (0)
Leptospirosis (Infections and infestations) | 1 (1) | 0 (0)
Liver Abscess (Infections and infestations) | 1 (1) | 0 (0)
Localised Infection (Infections and infestations) | 2 (2) | 0 (0)
Lung Abscess (Infections and infestations) | 1 (1) | 0 (0)
Lyme Disease (Infections and infestations) | 1 (1) | 0 (0)
Medical Device Site Joint Infection (Infections and infestations) | 3 (3) | 0 (0)
Meningitis Viral (Infections and infestations) | 1 (1) | 0 (0)
Meningoencephalitis Herpetic (Infections and infestations) | 1 (1) | 0 (0)
Muscle Abscess (Infections and infestations) | 1 (1) | 0 (0)
Necrotising Fasciitis (Infections and infestations) | 2 (2) | 0 (0)
Necrotising Soft Tissue Infection (Infections and infestations) | 1 (1) | 0 (0)
Ophthalmic Herpes Zoster (Infections and infestations) | 1 (1) | 0 (0)
Oral Candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 6 (6) | 1 (1)
Osteomyelitis Acute (Infections and infestations) | 1 (1) | 0 (0)
Pancreas Infection (Infections and infestations) | 2 (2) | 0 (0)
Pelvic Abscess (Infections and infestations) | 1 (1) | 0 (0)
Perineal Abscess (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 7 (7) | 0 (0)
Pneumonia (Infections and infestations) | 52 (55) | 1 (1)
Pneumonia Chlamydial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia Pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia Streptococcal (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia Viral (Infections and infestations) | 1 (1) | 0 (0)
Post Procedural Infection (Infections and infestations) | 1 (1) | 0 (0)
Postoperative Abscess (Infections and infestations) | 1 (1) | 0 (0)
Postoperative Wound Infection (Infections and infestations) | 2 (2) | 0 (0)
Psoas Abscess (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary Tuberculosis (Infections and infestations) | 2 (2) | 0 (0)
Pyelonephritis (Infections and infestations) | 3 (3) | 0 (0)
Pyelonephritis Acute (Infections and infestations) | 5 (7) | 0 (0)
Pyelonephritis Chronic (Infections and infestations) | 1 (1) | 0 (0)
Relapsing Fever (Infections and infestations) | 1 (1) | 0 (0)
Renal Abscess (Infections and infestations) | 1 (1) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Salmonellosis (Infections and infestations) | 1 (1) | 0 (0)
Salpingitis (Infections and infestations) | 1 (1) | 0 (0)
Salpingo-Oophoritis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 6 (6) | 0 (0)
Septic Arthritis Neisserial (Infections and infestations) | 1 (1) | 0 (0)
Septic Shock (Infections and infestations) | 6 (6) | 0 (0)
Sialoadenitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Soft Tissue Infection (Infections and infestations) | 3 (3) | 0 (0)
Staphylococcal Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal Infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal Skin Infection (Infections and infestations) | 2 (2) | 0 (0)
Subcutaneous Abscess (Infections and infestations) | 5 (5) | 0 (0)
Subdural Abscess (Infections and infestations) | 1 (1) | 0 (0)
Tooth Abscess (Infections and infestations) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 2 (2) | 0 (0)
Tubo-Ovarian Abscess (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 4 (4) | 0 (0)
Urosepsis (Infections and infestations) | 2 (2) | 0 (0)
Viral Myositis (Infections and infestations) | 1 (1) | 0 (0)
Wound Infection (Infections and infestations) | 2 (2) | 0 (0)
Wound Infection Staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Wound Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Abdominal Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Accidental Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alcohol Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anaemia Postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle Fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Comminuted Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dislocation Of Vertebra (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 8 (8) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 7 (7) | 1 (1)
Foot Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fractured Sacrum (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Gastrointestinal Stoma Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gun Shot Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip Fracture (Injury, poisoning and procedural complications) | 5 (5) | 0 (0)
Humerus Fracture (Injury, poisoning and procedural complications) | 5 (5) | 1 (1)
Incision Site Fibrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incisional Hernia (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint Dislocation (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Ligament Sprain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Multiple Injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Patella Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Pelvic Fracture (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Periorbital Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Periprosthetic Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Periprosthetic Osteolysis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post Procedural Fistula (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Procedural Shock (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 5 (5) | 0 (0)
Spinal Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural Haematoma (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Tendon Rupture (Injury, poisoning and procedural complications) | 5 (5) | 0 (0)
Thermal Burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia Fracture (Injury, poisoning and procedural complications) | 5 (5) | 0 (0)
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ulna Fracture (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 9 (9) | 0 (0)
Fungal Test Positive (Investigations) | 1 (1) | 0 (0)
Hiv Test False Positive (Investigations) | 1 (1) | 0 (0)
Neutrophil Count Decreased (Investigations) | 1 (1) | 0 (0)
Oxygen Saturation Decreased (Investigations) | 1 (1) | 0 (0)
Transaminases Increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemic Hyperosmolar Nonketotic Syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Latent Autoimmune Diabetes In Adults (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Ankle Deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 6 (9) | 0 (0)
Atlantoaxial Subluxation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Bone Cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Foot Deformity (Musculoskeletal and connective tissue disorders) | 14 (19) | 0 (0)
Hand Deformity (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Joint Destruction (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Knee Deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 45 (52) | 2 (2)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Osteoporotic Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 32 (33) | 1 (1)
Rheumatoid Nodule (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Wrist Deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma Of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ameloblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anal Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 0 (0)
Benign Neoplasm Of Thyroid Gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder Cancer Stage Ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Breast Cancer Stage Ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bronchial Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cervix Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Clear Cell Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Colorectal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Eye Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Fibroadenoma Of Breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gallbladder Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung Carcinoma Cell Type Unspecified Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian Germ Cell Teratoma Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Parathyroid Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pituitary Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pleomorphic Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Prostatic Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Refractory Anaemia With An Excess Of Blasts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Serous Cystadenocarcinoma Ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small Intestine Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous Cell Carcinoma Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous Cell Carcinoma Of The Cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Carpal Tunnel Syndrome (Nervous system disorders) | 4 (4) | 0 (0)
Cerebellar Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral Haematoma (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral Infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 5 (6) | 0 (0)
Cerebrovascular Insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
Depressed Level Of Consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 3 (3) | 0 (0)
Haemorrhage Intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic Stroke (Nervous system disorders) | 0 (0) | 2 (2)
Haemorrhagic Transformation Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Intraventricular Haemorrhage (Nervous system disorders) | 2 (2) | 0 (0)
Ischaemic Stroke (Nervous system disorders) | 2 (2) | 1 (1)
Lumbar Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Multifocal Motor Neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Partial Seizures (Nervous system disorders) | 2 (2) | 0 (0)
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 2 (2) | 0 (0)
Ruptured Cerebral Aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 0 (0)
Subarachnoid Haemorrhage (Nervous system disorders) | 3 (3) | 0 (0)
Syncope (Nervous system disorders) | 4 (4) | 0 (0)
Transient Global Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 6 (7) | 0 (0)
Vascular Headache (Nervous system disorders) | 1 (1) | 0 (0)
Abortion Missed (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Device Breakage (Product Issues) | 2 (4) | 0 (0)
Device Dislocation (Product Issues) | 1 (1) | 0 (0)
Device Loosening (Product Issues) | 1 (1) | 0 (0)
Device Malfunction (Product Issues) | 2 (2) | 0 (0)
Acute Psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol Abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Bipolar Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Conversion Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Major Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Mixed Anxiety And Depressive Disorder (Psychiatric disorders) | 1 (2) | 0 (0)
Paranoia (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide Attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 3 (3) | 0 (0)
Calculus Urinary (Renal and urinary disorders) | 0 (0) | 1 (1)
Cystitis Haemorrhagic (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 7 (7) | 0 (0)
Renal Colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0)
Urethral Stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Acquired Hydrocele (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Adnexa Uteri Cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast Enlargement (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast Hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cervical Dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cervical Polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Endometrial Hyperplasia (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Menometrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Ovarian Cyst (Reproductive system and breast disorders) | 4 (4) | 0 (0)
Pelvic Prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine Haemorrhage (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Uterine Prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial Hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diaphragmatic Abnormal Relaxation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Idiopathic Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pneumothorax Spontaneous (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 2 (3)
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cutaneous Lupus Erythematosus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin Necrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Subcutaneous Emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Toxic Skin Eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pregnancy Of Partner (Social circumstances) | 1 (1) | 0 (0)
Accelerated Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Aortic Embolus (Vascular disorders) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 8 (8) | 0 (0)
Haematoma (Vascular disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Hypertensive Crisis (Vascular disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 0 (0)
Hypovolaemic Shock (Vascular disorders) | 1 (1) | 0 (0)
Iliac Artery Embolism (Vascular disorders) | 1 (1) | 0 (0)
Pelvic Venous Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral Artery Occlusion (Vascular disorders) | 1 (2) | 0 (0)
Peripheral Embolism (Vascular disorders) | 1 (1) | 0 (0)
Peripheral Ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Peripheral Venous Disease (Vascular disorders) | 1 (1) | 0 (0)
Varicose Vein (Vascular disorders) | 3 (3) | 0 (0)
Venous Thrombosis Limb (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sarilumab + Disease Modifying Anti-Rheumatic Drugs (DMARD) (N=1910) | Sarilumab Monotherapy (N=111)
Leukopenia (Blood and lymphatic system disorders) | 101 (181) | 4 (5)
Neutropenia (Blood and lymphatic system disorders) | 348 (786) | 18 (64)
Diarrhoea (Gastrointestinal disorders) | 122 (153) | 2 (2)
Injection Site Erythema (General disorders) | 111 (751) | 0 (0)
Bronchitis (Infections and infestations) | 215 (301) | 12 (19)
Influenza (Infections and infestations) | 124 (160) | 3 (4)
Nasopharyngitis (Infections and infestations) | 249 (390) | 14 (26)
Pharyngitis (Infections and infestations) | 110 (129) | 4 (4)
Upper Respiratory Tract Infection (Infections and infestations) | 303 (574) | 16 (21)
Urinary Tract Infection (Infections and infestations) | 264 (428) | 14 (22)
Accidental Overdose (Injury, poisoning and procedural complications) | 330 (496) | 20 (22)
Fall (Injury, poisoning and procedural complications) | 109 (122) | 3 (3)
Alanine Aminotransferase Increased (Investigations) | 201 (287) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 87 (109) | 9 (11)
Back Pain (Musculoskeletal and connective tissue disorders) | 122 (141) | 6 (6)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 227 (357) | 16 (31)
Cough (Respiratory, thoracic and mediastinal disorders) | 62 (70) | 7 (7)
Hypertension (Vascular disorders) | 235 (271) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2015-08-31): https://cdn.clinicaltrials.gov/large-docs/52/NCT01146652/Prot_000.pdf
  • Statistical Analysis Plan (2015-12-22): https://cdn.clinicaltrials.gov/large-docs/52/NCT01146652/SAP_001.pdf